CLINICAL TRIAL: NCT01276639
Title: Phase 3 Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Of The Efficacy And Safety Of 2 Oral Doses Of CP-690,550 In Subjects With Moderate To Severe Chronic Plaque Psoriasis
Brief Title: A One-Year Study To Evaluate The Effects And Safety Of CP-690,550 In Patients With Moderate To Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921078
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Psoriasis
Keywords: Xeljanz; tofacitinib; chronic; Pruritus; Itch; DLQI; severe; moderate; treatment; safety; efficacy; CP-690,550; Plaque Psoriasis; Psoriasis Vulgaris; Jax-inhibitor; Oral Treatment
MeSH Terms: conditions — Psoriasis; Bronchiolitis Obliterans Syndrome; Pruritus; Lymphoma, Follicular | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active Treatment 10 mg BID (Experimental)
  Interventions: Drug: CP-690,550
- ActiveTreatment 5 mg BID (Experimental)
  Interventions: Drug: CP-690,550
- Placebo Treatment (Placebo Comparator)
  Interventions: Drug: Placebo/CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — 10 mg oral BID, Continuous treatment for 52 Weeks
  Arms: Active Treatment 10 mg BID
Drug: CP-690,550 — 5 mg oral BID, Continuous treatment for 52 Weeks
  Arms: ActiveTreatment 5 mg BID
Drug: Placebo/CP-690,550 — 0 mg oral BID, Continuous treatment for 16 Weeks; 10 mg oral BID, Continuous Treatment for 36 Weeks (after completion of 16 Weeks of Placebo)
  Arms: Placebo Treatment
Drug: Placebo/CP-690,550 — 0 mg oral BID, Continuous treatment for 16 Weeks; 5 mg oral BID, Continuous Treatment for 36 Weeks (after completion of 16 Weeks of Placebo)
  Arms: Placebo Treatment

SUMMARY:
The main objective of this study is to compare the effects of CP-690,550 with the effects of placebo in patients being treated for moderate to severe chronic plaque psoriasis. This one-year study will also evaluate the safety and tolerability of CP-690,550 versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years or older with diagnosis for at least 12 months of moderate to severe plaque psoriasis covering as least 10%of body surface area
* a Psoriasis Area and Severity Index (PASI) score of 12 and are considered to be candidates for systemic or light therapy
* No evidence of active or latent tuberculosis

Exclusion Criteria:

* Non-plaque or drug induced forms of psoriasis
* cannot discontinue current oral, injectible or topical therapy for psoriasis or cannot discontinue phototherapy (PUVA or UVB)
* any uncontrolled significant medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (74):
- United States (32):
  - Radiant Research, Inc., Birmingham, Alabama
  - University of California, Irvine - Dermatology Research, Irvine, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - The Savin Center, P.C., New Haven, Connecticut
  - Renstar Medical Research, Ocala, Florida
  - Academic Alliance in Dermatology, Tampa, Florida
  - Atlanta Dermatology, Vein & Research Center, P.C., Alpharetta, Georgia
  - Peachtree Dermatology Associates Research Center, Atlanta, Georgia
  - MedaPhase Inc., Newnan, Georgia
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital - Clinical Unit for Research Trials and Outcomes in Skin, Boston, Massachusetts
  - Skin Specialists, P.C., Omaha, Nebraska
  - New York University School of Medicine, New York, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - Raleigh Radiology Blue Ridge, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Central Sooner Research, Norman, Oklahoma
  - Baker Allergy, Asthma and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - University of Pittsburgh Medical Center - Department of Dermatology, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Dermatology Associates of Knoxville, PC, Knoxville, Tennessee
  - Modern Research Associates, PLLC, Dallas, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Rockwood Dermatology Center, Spokane, Washington
  - Rockwood Research Center, Spokane, Washington
  - Wenatchee Valley Medical Center - Clinical Research Department, Wenatchee, Washington
  - Madison Skin and Research, Inc., Madison, Wisconsin
- Canada (10):
  - Dermadvances Research, Winnipeg, Manitoba
  - Dr. Zohair Tomi PMC Inc., St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Research Associates Ltd., Halifax, Nova Scotia
  - Ultranova Skincare, Barrie, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Oakville Dermatology Laser Centre, Oakville, Ontario
  - Office of Dr. Michael Robern, Ottawa, Ontario
  - K.Papp Clinical Research Inc., Waterloo, Ontario
  - CRCMRGilbert Inc., Centre de Dermatologie Maizerets, Québec, Quebec
- Colombia (2):
  - Centro de Reumatologia y Ortopedia, Barranquilla, Atlántico
  - Riesgo de Fractura S.A, Bogot, Cundinamarca
- Germany (10):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Aerztehaus "Rudolf Virchow", Berlin
  - Klinik und Poliklinik fuer Dermatologie und Allergologie der Universitaet Bonn, Bonn
  - Universitaetsklinik Carl Gustav Carus, Dresden
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitaetsklinikum Muenster, Münster
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Praxisklinik fuer Dermatologie, Allergologie und Venenheilkunde, Vechta
  - Facharzt fuer Dermatologie und Venerologie, Allergologie, Wuppertal
- Hungary (3):
  - Bacs-Kiskun Megyei Onkormanyzat Korhaza Szegedi Tudomanyegyetem AOK Oktato Korhaza, Kecskemét
  - Josa Andras Oktatokorhaz, Borgyogyaszat, Nyíregyháza
  - Pecsi Tudomanyegyetem/Bor-, Nemikortani es Onkodermatologiai Klinika, Pécs
- Japan (5):
  - Gunma University Hospital, Maebashi, Gunma
  - JR Sapporo hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Chūōku, Kobe
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Social Insurance Chuo General Hospital, Shinjyuku-ku, Tokyo
- Centro de Dermatologia de Monterrey, Monterrey, Nuevo León, Mexico
- Poland (4):
  - Poznanski Osrodek Medyczny, Poznan
  - Katedra i Klinika Chorob Skornych i Wenerycznych, Pomorski Uniwersytet Medyczny, Szczecin
  - Katedra i Klinika Dermatologii, Wenerologii i Alergologii Akademii Medycznej we Wroclawiu, Wroclaw
  - Oddzial Dermatologiczny, Wroclaw
- Clinical Hospital Center Zvezdara, Belgrade, Serbia
- Taiwan (2):
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Ukraine (4):
  - Dept of Dermatology and Venerology of SI "Crimean State Medical University n.a. S.I. Georgiyevskyj", Simferopol, Autonomous Republic of Crimea
  - Dept of Dermatology, Infectious and Parasitic Skin Diseases, Kharkiv, Ukraine
  - Ternopil Regional Clinical Dermatovenerologic Dispensary, Ternopil, Ukraine
  - Dept of Dermatology and Venereology of National Medical University n.a. O.O. Bogomolets, Kyiv

REFERENCES:
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Wolk R, Armstrong EJ, Hansen PR, Thiers B, Lan S, Tallman AM, Kaur M, Tatulych S. Effect of tofacitinib on lipid levels and lipid-related parameters in patients with moderate to severe psoriasis. J Clin Lipidol. 2017 Sep-Oct;11(5):1243-1256. doi: 10.1016/j.jacl.2017.06.012. Epub 2017 Jun 24. PMID 28751001
- [Derived] Merola JF, Elewski B, Tatulych S, Lan S, Tallman A, Kaur M. Efficacy of tofacitinib for the treatment of nail psoriasis: Two 52-week, randomized, controlled phase 3 studies in patients with moderate-to-severe plaque psoriasis. J Am Acad Dermatol. 2017 Jul;77(1):79-87.e1. doi: 10.1016/j.jaad.2017.01.053. Epub 2017 Apr 7. PMID 28396102
- [Derived] Tan H, Valdez H, Griffins CE, Mrowietz U, Tallman A, Wolk R, Gordon K. Early clinical response to tofacitinib treatment as a predictor of subsequent efficacy: Results from two phase 3 studies of patients with moderate-to-severe plaque psoriasis. J Dermatolog Treat. 2017 Feb;28(1):3-7. doi: 10.1080/09546634.2016.1214671. Epub 2016 Aug 18. PMID 27538247
- [Derived] Papp KA, Menter MA, Abe M, Elewski B, Feldman SR, Gottlieb AB, Langley R, Luger T, Thaci D, Buonanno M, Gupta P, Proulx J, Lan S, Wolk R; OPT Pivotal 1 and OPT Pivotal 2 investigators. Tofacitinib, an oral Janus kinase inhibitor, for the treatment of chronic plaque psoriasis: results from two randomized, placebo-controlled, phase III trials. Br J Dermatol. 2015 Oct;173(4):949-61. doi: 10.1111/bjd.14018. PMID 26149717
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921078&StudyName=A%20One-Year%20Study%20To%20Evaluate%20The%20Effects%20And%20Safety%20Of%20CP-690%2C550%20In%20Patients%20With%20Moderate%20To%20Severe%20Chronic%20Plaque%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Outcome measures reporting results up to week 16 consist of single placebo arm as reporting group while outcome measures reporting results up to week 52 consist of 2 separate arms (for participants re-randomized at week 16 to receive CP-690,550 5 milligram [mg] or 10 mg).
Groups:
- CP-690,550 5 mg: CP-690,550 (tofacitinib) 5 milligram (mg) tablet orally twice daily up to Week 52.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily up to Week 52.
- Placebo: Placebo matched to CP-690,550 tablet orally twice daily up to Week 16. Participants in this group were re-randomized to CP-690,550 5 mg or CP-690,550 10 mg treatment at Week 16.
- Placebo, CP-690,550 5 mg: Participants who were re-assigned to this group from placebo at Week 16 and thereafter received CP-690,550 5 mg tablet orally twice daily up to Week 52.
- Placebo, CP-690,550 10 mg: Participants who were re-assigned to this group from placebo at Week 16 and thereafter received CP-690,550 10 mg tablet orally twice daily up to Week 52.
Period: Week 0 to 16
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Started | 363 | 361 | 177 | 0 | 0
Treated | 363 | 360 | 177 | 0 | 0
Completed | 313 | 320 | 132 | 0 | 0
Not Completed | 50 | 41 | 45 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 11 | 8 | 11 | 0 | 0
Not completed — Lack of Efficacy | 20 | 15 | 25 | 0 | 0
Not completed — Lost to Follow-up | 3 | 5 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 5 | 4 | 0 | 0
Not completed — Other | 7 | 7 | 2 | 0 | 0
Not completed — Randomized, But Not Treated | 0 | 1 | 0 | 0 | 0
Period: Week 16 to 52
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Started | 313 | 320 | 0 | 66 | 66
Completed | 186 | 219 | 0 | 50 | 45
Not Completed | 127 | 101 | 0 | 16 | 21
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 13 | 0 | 1 | 3
Not completed — Lack of Efficacy | 99 | 71 | 0 | 14 | 13
Not completed — Lost to Follow-up | 3 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 4 | 0 | 0 | 1
Not completed — Other | 10 | 12 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of investigational drug (CP-690,550 or placebo).
Groups:
- CP-690,550 5 mg: CP-690,550 5 mg tablet orally twice daily up to Week 52.
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Total
Number analyzed (Participants) | 363 | 360 | 177 | 900
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (13.4) | 45.2 (12.8) | 45.0 (12.6) | 45.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 99 | 56 | 257
  Male | 261 | 261 | 121 | 643

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Physician Global Assessment (PGA) of Psoriasis Score of 'Clear' or 'Almost Clear' at Week 16
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear).
Time Frame: Week 16
Population: Full analysis set (FAS) included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (CP-690,550 or placebo). Non-Responder Imputation (NRI) method (participants with missing values considered as non-responders) was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 363 | 360 | 177
percentage of participants | 41.87 | 59.17 | 9.04
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; For primary endpoint, step-down procedure used to preserve Type I error, sequential order of testing: PGA response for CP-690,550 10 mg versus (vs) placebo at Week 16; Psoriasis Area and Severity Index 75 (PASI75) response for CP-690,550 10 mg vs placebo at Week 16; PGA response for CP-690,550 5 mg vs placebo at Week 16; PASI75 response for CP-690,550 5 mg vs placebo at Week 16. If comparison at preceding step was significant, only then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel statistics adjusted for pooled investigator sites was used for the analysis. Each hypothesis was tested against placebo at significance level of 0.05 (2-sided); Odds Ratio (OR) = 6.46, 95% CI 2-sided [4.40 to 15.03]
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 12.45, 95% CI 2-sided [9.01 to 31.88]
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; Test type: Superiority or Other; p < 0.0001, Normal approximation; Percent difference = 17.29, 95% CI 2-sided [10.11 to 24.47], Standard Error of Mean 3.66

2. Primary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 75 (PASI 75) Response at Week 16
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 75 response was defined as at least a 75 percent (%) reduction in PASI relative to Baseline.
Time Frame: Week 16
Population: FAS included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (CP-690,550 or placebo). NRI method (participants with missing values considered as non-responders) was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 363 | 360 | 177
percentage of participants | 39.94 | 59.17 | 6.21
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 8.93, 95% CI 2-sided [5.25 to 21.84]
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 20.81, 95% CI 2-sided [11.90 to 49.86]
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; Test type: Superiority or Other; p < 0.0001, Normal approximation; Percent difference = 19.22, 95% CI 2-sided [12.07 to 26.37], Standard Error of Mean 3.65

3. Secondary Outcome: Percent Change From Baseline in Total Body Surface Area (BSA) With Psoriasis at Week 16
Description: Assessment of BSA with psoriasis was estimated by means of the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumb together) represented approximately 1% of the total BSA. Body regions are assigned specific number of handprints with percentage [Head and neck = 10% (10 handprints), upper extremities = 20% (20 handprints), Trunk (including axillae and groin) = 30% (30 handprints), lower extremities (including buttocks) = 40% (40 handprints)]. The number of handprints of psoriatic skin in a body region was used to determine the extent (%) to which a body region was involved with psoriasis. The total BSA affected was the summation of individual regions affected.
Time Frame: Baseline, Week 16
Population: FAS included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (CP-690,550 or placebo). Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 359 | 358 | 177
percent change | -51.94 (2.45) | -67.20 (2.44) | 1.62 (3.59)
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; For key secondary endpoint, family-wise step-down procedure was used to control Type I error. Sequential order of testing: percent change in BSA at Week 16,PASI90 response at Week 16, change in Dermatology Life Quality Index(DLQI) total score at Week 16,PGA response at Week 4,PASI75 at Week 4, change in DLQI total score at Week 4, percent change in Nail Psoriasis Severity Index(NAPSI) score at Week 16. If comparison at preceding step was significant, then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Mixed model analysis with fixed effects for treatment, visit, treatment-by-visit interaction,baseline value and repeated measures for visit. Unstructured covariance matrix was used. Each hypothesis was tested at significance level of 0.025 (2-sided); Least squares (LS) mean difference = -53.56, 95% CI 2-sided [-62.08 to -45.04], Standard Error of Mean 4.34
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -68.82, 95% CI 2-sided [-77.33 to -60.31], Standard Error of Mean 4.34
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; LS mean difference was derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction, baseline value and repeated measures for visit. Unstructured covariance matrix was used; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS mean difference = -15.26, 95% CI 2-sided [-22.04 to -8.48], Standard Error of Mean 3.46

4. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 90 (PASI 90) Response at Week 16
Description: The PASI quantifies the severity of a participant's psoriasis based on both, lesion severity and the percent of BSA affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 90 response was defined as at least a 90% reduction in PASI relative to Baseline.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 363 | 360 | 177
percentage of participants | 19.83 | 39.44 | 0.56
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; For key secondary endpoint, family-wise step-down procedure was used to control Type I error. Sequential order of testing: percent change in BSA at Week 16, PASI90 response at Week 16, change in DLQI total score at Week 16, PGA response at Week 4, PASI75 response at Week 4, change in DLQI total score at Week 4, percent change in NAPSI score at Week 16. If comparison at preceding step was significant, then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel statistics adjusted for pooled investigator sites was used for the analysis. Each hypothesis was tested at significance level of 0.025 (2-sided); Odds Ratio (OR) = 34.55, 95% CI 2-sided [7.46 to 1786.9]
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 98.05, 95% CI 2-sided [23.49 to 5689.8]
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; Test type: Superiority or Other; p < 0.0001, Normal approximation; Percent difference = 19.61, 95% CI 2-sided [13.10 to 26.11], Standard Error of Mean 3.32

5. Secondary Outcome: Dermatology Life Quality Index (DLQI) Total Score
Description: The DLQI is a 10 item general dermatology questionnaire that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI item response options are rated by the participant from 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life.
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 363 | 359 | 177
units on a scale | 12.46 (6.89) | 12.87 (6.91) | 14.01 (7.06)

6. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 4 and 16
Description: as for outcome 5
Time Frame: Week 4, 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 358 | 357 | 177
units on a scale
  Change at Week 4 | -5.59 (0.25) | -6.40 (0.25) | -1.69 (0.35)
  Change at Week 16 | -6.91 (0.30) | -8.90 (0.29) | -1.93 (0.44)
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; Week4: For key secondary endpoint, family-wise step-down procedure was used to control Type I error. Sequential order of testing: percent change in BSA at Week 16, PASI90 response at Week 16, change in DLQI total score at Week 16, PGA response at Week 4, PASI75 response at Week 4, change in DLQI total score at Week 4, percent change in NAPSI score at Week 16. If comparison at preceding step was significant, then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -3.90, 95% CI 2-sided [-4.75 to -3.05], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; Week 4: For key secondary endpoint, family-wise step-down procedure was used to control Type I error. Sequential order of testing: percent change in BSA at Week 16, PASI90 response at Week 16, change in DLQI total score at Week 16, PGA response at Week 4, PASI75 response at Week 4, change in DLQI total score at Week 4, percent change in NAPSI score at Week 16. If comparison at preceding step was significant, then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -4.71, 95% CI 2-sided [-5.56 to -3.86], Standard Error of Mean 0.43
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; Week 4: LS mean difference was derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction, baseline value and repeated measures for visit. Unstructured covariance matrix was used; Test type: Superiority or Other; p = 0.0212, Mixed Models Analysis; LS mean difference = -0.81, 95% CI 2-sided [-1.50 to -0.12], Standard Error of Mean 0.35
Statistical Analysis 4: Comparison: CP-690,550 5 mg vs Placebo; Week 16: For key secondary endpoint, family-wise step-down procedure was used to control Type I error. Sequential order of testing: percent change in BSA at Week 16, PASI90 response at Week 16, change in DLQI total score at Week 16, PGA response at Week 4, PASI75 response at Week 4, change in DLQI total score at Week 4, percent change in NAPSI score at Week 16. If comparison at preceding step was significant, then subsequent comparisons were significant; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -4.98, 95% CI 2-sided [-6.02 to -3.95], Standard Error of Mean 0.53
Statistical Analysis 5: Comparison: CP-690,550 10 mg vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -6.97, 95% CI 2-sided [-8.00 to -5.94], Standard Error of Mean 0.53
Statistical Analysis 6: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; Week 16: LS mean difference was derived from mixed model with fixed effects for treatment, visit, treatment-by-visit interaction, baseline value and repeated measures for visit. Unstructured covariance matrix was used; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS mean difference = -1.99, 95% CI 2-sided [-2.80 to -1.17], Standard Error of Mean 0.42

7. Secondary Outcome: Percentage of Participants With Physician Global Assessment (PGA) of Psoriasis Score of 'Clear' or 'Almost Clear' at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 363 | 360 | 177
percentage of participants | 17.08 | 23.06 | 2.26
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 8.34, 95% CI 2-sided [3.23 to 35.12]
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 11.53, 95% CI 2-sided [5.06 to 54.42]
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; Test type: Superiority or Other; p = 0.0443, Normal approximation; Percent difference = 5.98, 95% CI 2-sided [0.15 to 11.80], Standard Error of Mean 2.97

8. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 75 (PASI 75) Response at Week 4
Description: The PASI quantifies the severity of a participant's psoriasis based on both, lesion severity and the percent of BSA affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 75 response was defined as at least 75% reduction in PASI relative to Baseline.
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 363 | 360 | 177
percentage of participants | 10.47 | 15.56 | 1.69
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 6.76, 95% CI 2-sided [2.11 to 35.77]
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 11.55, 95% CI 2-sided [3.64 to 59.98]
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; Test type: Superiority or Other; p = 0.0415, Normal approximation; Percent difference = 5.09, 95% CI 2-sided [0.19 to 9.98], Standard Error of Mean 2.50

9. Secondary Outcome: Percent Change From Baseline in Nail Psoriasis Severity Index (NAPSI) at Week 16
Description: The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each finger nail divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores = more severe psoriasis.
Time Frame: Baseline, Week 16
Population: FAS included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (CP-690,550 or placebo). Here 'N' (number of participants analyzed) signifies those participants who were evaluable (had nail psoriasis at Baseline and had at least one measurement during follow up) for this measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 237 | 242 | 102
percent change | -14.15 (9.47) | -41.48 (9.22) | 55.55 (14.84)
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -69.70, 95% CI 2-sided [-104.27 to -35.13], Standard Error of Mean 17.60
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -97.03, 95% CI 2-sided [-131.35 to -62.72], Standard Error of Mean 17.47
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.0391, Mixed Models Analysis; LS mean difference = -27.33, 95% CI 2-sided [-53.29 to -1.37], Standard Error of Mean 13.22

10. Secondary Outcome: Percent Probability of Participants Maintaining Physician Global Assessment (PGA) of Psoriasis Score of 'Clear' or 'Almost Clear' at Week 52
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). Maintenance of PGA response at Week 52 among participants achieving PGA response at Week 16 is reported. Percent probability and 95% confidence interval (CI) were estimated based on the product limit estimator in survival analyses. Event is loss of response. Probability of maintaining response is (1-probability of loss of response).
Time Frame: Week 52
Population: FAS participants who had PGA response at Week 16. Data was not analyzed for participants initially randomized to placebo arm as they were re-randomized to active treatment group at Week 16 and thus maintaining response at Week 52 was not relevant. 'N' (number of participants analyzed) = participants with non-missing post-baseline response data.
Measure: Number (95% Confidence Interval); unit: percent probability of response
Groups:
- CP-690,550 5 mg: Participants who received CP-690,550 5 mg tablet orally twice daily up to Week 52.
- CP-690,550 10 mg: Participants who received CP-690,550 10 mg tablet orally twice daily up to Week 52.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg
Number analyzed (Participants) | 151 | 209
percent probability of response | 60.17 [51.80 to 67.56] | 71.56 [64.81 to 77.24]

11. Secondary Outcome: Percent Probability of Participants Maintaining Psoriasis Area and Severity Index 75 (PASI 75) Response at Week 52
Description: The PASI quantifies severity of a participant's psoriasis based on both, lesion severity and percent of BSA affected. PASI is a composite scoring by investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 75 response = at least 75% reduction in PASI relative to Baseline. Maintenance of PASI 75 response at Week 52 among participants achieving PASI 75 response at Week 16 is reported. Percent probability and 95% CI were estimated based on the product limit estimator in survival analyses. Event is loss of response. Probability of maintaining response is (1-probability of loss of response).
Time Frame: Week 52
Population: FAS participants who had PASI 75 response at Week 16. Data was not analyzed for participants initially randomized to placebo arm as they were re-randomized to active treatment group at Week 16 and thus maintaining response at Week 52 was not relevant. 'N' (number of participants analyzed) = participants with non-missing post-baseline response data.
Measure: Number (95% Confidence Interval); unit: percent probability of response
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg
Number analyzed (Participants) | 145 | 209
percent probability of response | 73.75 [65.47 to 80.33] | 79.94 [73.75 to 84.82]

12. Secondary Outcome: Percent Probability of Participants Maintaining Psoriasis Area and Severity Index 90 (PASI 90) Response at Week 52
Description: The PASI quantifies severity of a participant's psoriasis based on both, lesion severity and percent of BSA affected. PASI is a composite scoring by investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 90 response = at least 90% reduction in PASI relative to Baseline. Maintenance of PASI 90 response at Week 52 among participants achieving PASI 90 response at Week 16 is reported. Percent probability and 95% CI were estimated based on the product limit estimator in survival analyses. Event is loss of response. Probability of maintaining response is (1-probability of loss of response).
Time Frame: Week 52
Population: FAS participants who had PASI 90 response at Week 16. Data was not analyzed for participants initially randomized to placebo arm as they were re-randomized to active treatment group at Week 16 and thus maintaining response at Week 52 was not relevant. 'N' (number of participants analyzed) = participants with non-missing post-baseline response data.
Measure: Number (95% Confidence Interval); unit: percent probability of response
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg
Number analyzed (Participants) | 72 | 140
percent probability of response | 61.79 [49.37 to 72.01] | 70.58 [62.12 to 77.49]

13. Secondary Outcome: Time to Achieve a Physician Global Assessment (PGA) of Psoriasis Score of 'Clear' or 'Almost Clear'
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). Median time to achieve a PGA response up to week 16 is reported. The median time to event was estimated based on the probability of event-rate based on life table estimates (not the observed rate as in outcome measure 1). Median time to event is not estimable if the estimated probability of response by Week 16 is less than 50%.
Time Frame: Baseline up to Week 16
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 359 | 358 | 177
weeks | 16.0 [12.0 to NA] — Upper limit was not estimable based on the log-log transformation method. | 12.0 [8.0 to 12.0] | NA [NA to NA] — Data was not estimable because estimated probability of response by Week 16 was less than 50%.
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; Test type: Superiority or Other; p < 0.0001, Log Rank

14. Secondary Outcome: Time to Achieve Psoriasis Area and Severity Index 75 (PASI 75) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 75 response was defined as at least 75% reduction in PASI relative to Baseline. The median time to event was estimated based on the probability of event-rate based on life table estimates (not the observed rate as in outcome measure 2). Median time to event is not estimable if the estimated probability of response by Week 16 is less than 50%.
Time Frame: Baseline up to Week 16
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 359 | 358 | 177
weeks | NA [16.0 to NA] — Data was not estimable because estimated probability of response by Week 16 was less than 50%. | 12.0 [NA to NA] — Upper and lower limits were not estimable based on the log-log transformation method. | NA [NA to NA] — Data was not estimable because estimated probability of response by Week 16 was less than 50%.
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; Test type: Superiority or Other; p < 0.0001, Log Rank

15. Secondary Outcome: Time to Achieve Psoriasis Area and Severity Index 50 (PASI 50) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 50 response was defined as at least 50% reduction in PASI relative to Baseline. The median time to event was estimated based on the probability of event-rate based on life table estimates (not the observed rate as in outcome measure 26). Median time to event is not estimable if the estimated probability of response by Week 16 is less than 50%.
Time Frame: Baseline up to Week 16
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 359 | 358 | 177
weeks | 8.0 [8.0 to 12.0] | 8.0 [NA to NA] — Upper and lower limits were not estimable based on the log-log transformation method. | NA [NA to NA] — Data was not estimable because estimated probability of response by Week 16 was less than 50%.
Statistical Analysis 1: Comparison: CP-690,550 5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: CP-690,550 10 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 3: Comparison: CP-690,550 5 mg vs CP-690,550 10 mg; Test type: Superiority or Other; p < 0.0001, Log Rank

16. Secondary Outcome: Percentage of Participants With Physician Global Assessment (PGA) of Psoriasis Score of 'Clear' or 'Almost Clear'
Description: as for outcome 1
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: FAS: all randomized participants who received at least 1 dose of the randomized investigational drug (CP-690,550 or placebo). Analysis population for "Placebo, CP-690,550" groups included FAS participants who were re-randomized at Week 16 to receive CP-690,550 5 mg or 10 mg. NRI method was used to impute missing values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
percentage of participants
  Week 2 | 5.23 [2.94 to 7.53] | 10.00 [6.90 to 13.10] | 3.03 [0.00 to 7.17] | 0.00 [0.00 to 0.00]
  Week 4 | 17.08 [13.21 to 20.95] | 23.06 [18.70 to 27.41] | 6.06 [0.30 to 11.82] | 0.00 [0.00 to 0.00]
  Week 8 | 31.40 [26.63 to 36.18] | 46.39 [41.24 to 51.54] | 9.09 [2.16 to 16.03] | 6.06 [0.30 to 11.82]
  Week 12 | 37.74 [32.75 to 42.73] | 56.67 [51.55 to 61.79] | 12.12 [4.25 to 20.00] | 9.09 [2.16 to 16.03]
  Week 16 | 41.87 [36.80 to 46.95] | 59.17 [54.09 to 64.24] | 13.64 [5.36 to 21.92] | 10.61 [3.18 to 18.03]
  Week 20 | 45.45 [40.33 to 50.58] | 56.67 [51.55 to 61.79] | 39.39 [27.61 to 51.18] | 30.30 [19.22 to 41.39]
  Week 28 | 48.76 [43.62 to 53.90] | 62.22 [57.21 to 67.23] | 66.67 [55.29 to 78.04] | 65.15 [53.66 to 76.65]
  Week 40 | 42.70 [37.61 to 47.79] | 53.06 [47.90 to 58.21] | 53.03 [40.99 to 65.07] | 63.64 [52.03 to 75.24]
  Week 52 | 35.54 [30.61 to 40.46] | 46.67 [41.51 to 51.82] | 43.94 [31.97 to 55.91] | 59.09 [47.23 to 70.95]

17. Secondary Outcome: Percentage of Participants With Physician Global Assessment (PGA) of Psoriasis Score
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). Percentage of participants with each PGA score is reported.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: FAS. Analysis population for "Placebo, CP-690,550" groups included FAS participants who were re-randomized at Week 16 to receive CP-690,550 5 mg or 10 mg. NRI method was used to impute missing values. Here 'n' signifies those participants who were evaluable for this measure at specified time point for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
percentage of participants
  Baseline: Clear (n = 363, 360, 66, 66) | 0.00 | 0.00 | 0.00 | 0.00
  Baseline: Almost Clear (n = 363, 360, 66, 66) | 0.00 | 0.00 | 0.00 | 0.00
  Baseline: Mild (n = 363, 360, 66, 66) | 0.3 | 0.3 | 0.00 | 0.00
  Baseline: Moderate (n = 363, 360, 66, 66) | 88.2 | 88.9 | 97.0 | 92.4
  Baseline: Severe (n = 363, 360, 66, 66) | 11.6 | 10.8 | 3.0 | 7.6
  Week 2: Clear (n = 358, 358, 66, 64) | 0.00 | 0.00 | 0.00 | 0.00
  Week 2: Almost Clear (n = 358, 358, 66, 64) | 5.3 | 10.1 | 3.0 | 0.00
  Week 2: Mild (n = 358, 358, 66, 64) | 32.7 | 38.8 | 30.3 | 18.8
  Week 2: Moderate (n = 358, 358, 66, 64) | 57.0 | 46.1 | 63.6 | 70.3
  Week 2: Severe (n = 358, 358, 66, 64) | 5.0 | 5.0 | 3.0 | 10.9
  Week 4: Clear (n = 352, 350, 65, 66) | 1.4 | 3.4 | 0.00 | 0.00
  Week 4: Almost Clear (n = 352, 350, 65, 66) | 16.2 | 20.3 | 6.2 | 0.00
  Week 4: Mild (n = 352, 350, 65, 66) | 43.8 | 45.4 | 33.8 | 21.2
  Week 4: Moderate (n = 352, 350, 65, 66) | 35.5 | 28.3 | 55.4 | 71.2
  Week 4: Severe (n = 352, 350, 65, 66) | 3.1 | 2.6 | 4.6 | 7.6
  Week 8: Clear (n = 347, 350, 65, 66) | 3.7 | 10.6 | 0.00 | 0.00
  Week 8: Almost Clear (n = 347, 350, 65, 66) | 29.1 | 37.1 | 9.2 | 6.1
  Week 8: Mild (n = 347, 350, 65, 66) | 40.3 | 36.0 | 33.8 | 24.2
  Week 8: Moderate (n = 347, 350, 65, 66) | 24.2 | 14.6 | 53.8 | 65.2
  Week 8: Severe (n = 347, 350, 65, 66) | 2.6 | 1.7 | 3.1 | 4.5
  Week 12: Clear (n = 345, 345, 65, 66) | 7.8 | 17.4 | 1.5 | 0.00
  Week 12: Almost Clear (n = 345, 345, 65, 66) | 31.9 | 41.7 | 10.8 | 9.1
  Week 12: Mild (n = 345, 345, 65, 66) | 38.0 | 26.1 | 43.1 | 25.8
  Week 12: Moderate (n = 345, 345, 65, 66) | 19.4 | 13.0 | 41.5 | 54.5
  Week 12: Severe (n = 345, 345, 65, 66) | 2.9 | 1.7 | 3.1 | 10.6
  Week 16: Clear (n = 323, 335, 66, 66) | 12.1 | 25.7 | 0.00 | 3.0
  Week 16: Almost Clear (n = 323, 335, 66, 66) | 35.0 | 37.9 | 13.6 | 7.6
  Week 16: Mild (n = 323, 335, 66, 66) | 32.8 | 23.6 | 47.0 | 21.2
  Week 16: Moderate (n = 323, 335, 66, 66) | 17.6 | 11.3 | 34.8 | 62.1
  Week 16: Severe (n = 323, 335, 66, 66) | 2.5 | 1.5 | 4.5 | 6.1
  Week 20: Clear (n = 312, 321, 66, 65) | 16.3 | 31.2 | 7.6 | 9.2
  Week 20: Almost Clear (n = 312, 321, 66, 65) | 36.5 | 32.4 | 31.8 | 21.5
  Week 20: Mild (n = 312, 321, 66, 65) | 31.7 | 24.3 | 53.0 | 43.1
  Week 20: Moderate (n = 312, 321, 66, 65) | 14.7 | 11.5 | 7.6 | 23.1
  Week 20: Severe (n = 312, 321, 66, 65) | 0.6 | 0.6 | 0.00 | 3.1
  Week 28: Clear (n = 300, 307, 61, 61) | 23.3 | 34.2 | 14.8 | 29.5
  Week 28: Almost Clear (n = 300, 307, 61, 61) | 35.7 | 38.8 | 57.4 | 41.0
  Week 28: Mild (n = 300, 307, 61, 61) | 25.7 | 17.6 | 23.0 | 19.7
  Week 28: Moderate (n = 300, 307, 61, 61) | 14.3 | 8.8 | 4.9 | 6.6
  Week 28: Severe (n = 300, 307, 61, 61) | 1.0 | 0.7 | 0.00 | 3.3
  Week 40: Clear (n = 203, 242, 53, 57) | 35.5 | 45.9 | 18.9 | 55.3
  Week 40: Almost Clear (n = 203, 242, 53, 57) | 40.9 | 33.1 | 47.2 | 34.0
  Week 40: Mild (n = 203, 242, 53, 57) | 18.2 | 15.3 | 26.4 | 8.5
  Week 40: Moderate (n = 203, 242, 53, 57) | 4.9 | 5.4 | 7.5 | 2.1
  Week 40: Severe (n = 203, 242, 53, 57) | 0.5 | 0.4 | 0.00 | 0.00
  Week 52: Clear (n = 180, 219, 47, 46) | 31.7 | 43.4 | 19.1 | 54.3
  Week 52: Almost Clear (n = 180, 219, 47, 46) | 40.0 | 33.3 | 42.6 | 30.4
  Week 52: Mild (n = 180, 219, 47, 46) | 19.4 | 19.6 | 36.2 | 15.2
  Week 52: Moderate (n = 180, 219, 47, 46) | 8.9 | 3.7 | 2.1 | 0.00
  Week 52: Severe (n = 180, 219, 47, 46) | 0.00 | 0.00 | 0.00 | 0.00

18. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index 75 (PASI 75) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 75 response was defined as at least 75% reduction in PASI relative to Baseline. Percentage of participants with PASI 75 response is reported.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
percentage of participants
  Week 2 | 1.38 [0.18 to 2.58] | 2.22 [0.70 to 3.74] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 4 | 10.47 [7.32 to 13.62] | 15.56 [11.81 to 19.30] | 4.55 [0.00 to 9.57] | 0.00 [0.00 to 0.00]
  Week 8 | 23.69 [19.32 to 28.07] | 36.67 [31.69 to 41.64] | 6.06 [0.30 to 11.82] | 0.00 [0.00 to 0.00]
  Week 12 | 35.54 [30.61 to 40.46] | 55.28 [50.14 to 60.41] | 6.06 [0.30 to 11.82] | 7.58 [1.19 to 13.96]
  Week 16 | 39.94 [34.91 to 44.98] | 59.17 [54.09 to 64.24] | 9.09 [2.16 to 16.03] | 7.58 [1.19 to 13.96]
  Week 20 | 45.18 [40.06 to 50.30] | 59.44 [54.37 to 64.52] | 31.82 [20.58 to 43.06] | 24.24 [13.90 to 34.58]
  Week 28 | 49.86 [44.72 to 55.01] | 63.06 [58.07 to 68.04] | 59.09 [47.23 to 70.95] | 68.18 [56.94 to 79.42]
  Week 40 | 45.45 [40.33 to 50.58] | 56.94 [51.83 to 62.06] | 65.15 [53.66 to 76.65] | 68.18 [56.94 to 79.42]
  Week 52 | 38.84 [33.83 to 43.86] | 51.39 [46.23 to 56.55] | 54.55 [42.53 to 66.56] | 65.15 [53.66 to 76.65]

19. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: FAS. Analysis population for "Placebo, CP-690,550" groups included FAS participants who were re-randomized at Week 16 to receive CP-690,550 5 mg or 10 mg. Here 'n' signifies those participants who were evaluable for this measure at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
units on a scale
  Baseline (n=363,360,66,66) | 21.95 (8.99) | 22.73 (8.82) | 21.19 (8.54) | 23.03 (8.66)
  Week 2 (n=358,358,66,64) | 18.28 (9.63) | 17.30 (9.06) | 19.81 (10.28) | 22.11 (9.84)
  Week 4 (n=352,350,65,66) | 14.39 (8.75) | 13.10 (8.90) | 18.36 (10.86) | 20.63 (9.26)
  Week 8 (n=347,350,65,66) | 11.41 (9.08) | 8.97 (8.00) | 17.17 (10.32) | 20.13 (10.15)
  Week 12 (n=345,345,65,66) | 9.85 (9.38) | 6.94 (7.59) | 16.52 (10.45) | 19.38 (10.07)
  Week 16 (n=323,335,66,66) | 8.42 (9.05) | 5.74 (7.21) | 16.08 (10.41) | 19.71 (11.25)
  Week 20 (n=312,321,66,65) | 6.82 (7.23) | 4.95 (6.30) | 9.18 (7.21) | 11.79 (8.38)
  Week 28 (n=300,307,61,61) | 5.80 (6.87) | 4.01 (5.28) | 5.20 (5.95) | 5.23 (6.42)
  Week 40 (n=203,242,53,47) | 3.05 (3.71) | 2.64 (3.85) | 3.22 (3.70) | 1.64 (2.27)
  Week 52 (n=180,219,47,46) | 3.28 (3.71) | 2.47 (3.21) | 3.16 (3.22) | 1.64 (2.01)

20. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 2, 4, 8, 12, 16, 20, 28, 40 and 52
Description: as for outcome 19
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: FAS. Analysis population for "Placebo, CP-690,550" groups included FAS participants who were re-randomized at Week 16 to receive CP-690,550 5 mg or 10 mg. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 359 | 358 | 66 | 66
units on a scale
  Change at Week 2 | -3.87 (0.29) | -5.31 (0.29) | -1.79 (0.66) | -0.81 (0.67)
  Change at Week 4 | -7.61 (0.35) | -9.48 (0.35) | -3.14 (0.81) | -2.18 (0.81)
  Change at Week 8 | -10.61 (0.41) | -13.58 (0.41) | -4.45 (0.95) | -2.68 (0.95)
  Change at Week 12 | -12.02 (0.44) | -15.62 (0.44) | -4.97 (1.02) | -3.43 (1.02)
  Change at Week 16 | -12.90 (0.48) | -16.55 (0.48) | -5.51 (1.09) | -3.10 (1.09)
  Change at Week 20 | -14.36 (0.44) | -17.11 (0.44) | -12.41 (1.00) | -11.18 (1.00)
  Change at Week 28 | -15.53 (0.44) | -18.02 (0.43) | -16.21 (0.98) | -17.63 (0.98)
  Change at Week 40 | -15.15 (0.47) | -17.51 (0.46) | -16.16 (1.03) | -18.54 (1.05)
  Change at Week 52 | -14.70 (0.48) | -17.16 (0.47) | -15.69 (1.04) | -18.62 (1.06)

21. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Component Scores
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of BSA" affected. Basic characteristics of psoriatic lesions: erythema, induration, and scaling (PASI components) are scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]) according to a 5-point scale: 0 (no involvement); 1 (slight); 2 (moderate); 3 (marked); 4 (very marked). PASI component score range from 0 to 4, where higher scores indicate greater severity of psoriatic lesions.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
units on a scale
  Baseline: Erythema (Head\Neck) (n=363,360,66,66) | 2.31 (0.99) | 2.23 (1.01) | 2.38 (0.99) | 2.26 (0.90)
  Baseline: Erythema (Upper Limbs) (n=363,360,66,66) | 2.87 (0.64) | 2.88 (0.64) | 2.83 (0.54) | 2.92 (0.54)
  Baseline: Erythema (Trunk) (n=363,360,66,66) | 2.85 (0.77) | 2.91 (0.73) | 2.79 (0.85) | 3.08 (0.56)
  Baseline: Erythema (Lower Limbs) (n=363,360,66,66) | 3.21 (0.60) | 3.19 (0.62) | 3.14 (0.58) | 3.27 (0.62)
  Baseline: Induration (Head\Neck) (n=363,360,66,66) | 2.08 (0.97) | 1.96 (1.01) | 2.14 (0.97) | 2.02 (0.90)
  Baseline:Induration (Upper Limbs)(n=363,360,66,66) | 2.69 (0.71) | 2.65 (0.67) | 2.71 (0.58) | 2.68 (0.59)
  Baseline: Induration (Trunk) (n=363,360,66,66) | 2.60 (0.80) | 2.63 (0.77) | 2.53 (0.83) | 2.71 (0.78)
  Baseline:Induration (Lower Limbs)(n=363,360,66,66) | 2.91 (0.69) | 2.90 (0.66) | 2.83 (0.69) | 2.98 (0.69)
  Baseline: Scaling (Head\Neck) (n=363,360,66,66) | 2.32 (1.05) | 2.23 (1.08) | 2.33 (1.10) | 2.24 (1.07)
  Baseline: Scaling (Upper Limbs) (n=363,360,66,66) | 2.75 (0.78) | 2.71 (0.75) | 2.55 (0.59) | 2.76 (0.70)
  Baseline: Scaling (Trunk) (n=363,360,66,66) | 2.60 (0.86) | 2.60 (0.83) | 2.36 (0.82) | 2.77 (0.86)
  Baseline: Scaling (Lower Limbs) (n=363,360,66,66) | 2.98 (0.72) | 2.91 (0.72) | 2.77 (0.72) | 2.97 (0.78)
  Week 2: Erythema (Head\Neck) (n=358,358,66,64) | 1.84 (1.05) | 1.72 (1.05) | 2.14 (0.99) | 2.17 (0.88)
  Week 2: Erythema (Upper Limbs) (n=358,358,66,64) | 2.40 (0.80) | 2.26 (0.86) | 2.64 (0.62) | 2.83 (0.68)
  Week 2: Erythema (Trunk) (n=358,358,66,64) | 2.39 (0.92) | 2.28 (0.89) | 2.58 (0.88) | 2.91 (0.73)
  Week 2: Erythema (Lower Limbs) (n=358,358,66,64) | 2.75 (0.81) | 2.60 (0.83) | 2.98 (0.64) | 3.14 (0.69)
  Week 2: Induration (Head\Neck) (n=358,358,66,64) | 1.70 (1.05) | 1.48 (1.03) | 1.94 (0.99) | 1.92 (0.95)
  Week 2: Induration (Upper Limbs) (n=358,358,66,64) | 2.27 (0.83) | 2.11 (0.86) | 2.36 (0.76) | 2.58 (0.71)
  Week 2: Induration (Trunk) (n=358,358,66,64) | 2.20 (0.90) | 2.10 (0.92) | 2.32 (0.90) | 2.58 (0.75)
  Week 2: Induration (Lower Limbs) (n=358,358,66,64) | 2.50 (0.82) | 2.38 (0.84) | 2.62 (0.80) | 2.72 (0.74)
  Week 2: Scaling (Head\Neck) (n=358,358,66,64) | 1.85 (1.11) | 1.67 (1.11) | 2.03 (1.07) | 2.08 (1.13)
  Week 2: Scaling (Upper Limbs) (n=358,358,66,64) | 2.29 (0.93) | 2.08 (0.91) | 2.26 (0.75) | 2.58 (0.87)
  Week 2: Scaling (Trunk) (n=358,358,66,64) | 2.12 (1.00) | 2.00 (1.00) | 2.14 (1.04) | 2.50 (0.99)
  Week 2: Scaling (Lower Limbs) (n=358,358,66,64) | 2.50 (0.91) | 2.33 (0.92) | 2.53 (0.85) | 2.75 (0.82)
  Week 4: Erythema (Head\Neck) (n=352,350,65,66) | 1.45 (1.03) | 1.33 (1.06) | 1.89 (1.11) | 1.92 (0.97)
  Week 4: Erythema (Upper Limbs) (n=352,350,65,66) | 2.00 (0.88) | 1.85 (0.90) | 2.42 (0.81) | 2.73 (0.69)
  Week 4: Erythema (Trunk) (n=352,350,65,66) | 1.99 (0.99) | 1.83 (1.00) | 2.42 (0.97) | 2.74 (0.69)
  Week 4: Erythema (Lower Limbs) (n=352,350,65,66) | 2.35 (0.90) | 2.15 (0.91) | 2.78 (0.78) | 2.97 (0.68)
  Week 4: Induration (Head\Neck) (n=352,350,65,66) | 1.28 (0.98) | 1.11 (0.99) | 1.74 (1.06) | 1.74 (1.03)
  Week 4: Induration (Upper Limbs) (n=352,350,65,66) | 1.87 (0.90) | 1.73 (0.91) | 2.25 (0.83) | 2.53 (0.79)
  Week 4: Induration (Trunk) (n=352,350,65,66) | 1.80 (0.95) | 1.66 (1.00) | 2.15 (1.03) | 2.53 (0.81)
  Week 4: Induration (Lower Limbs) (n=352,350,65,66) | 2.06 (0.90) | 1.93 (0.92) | 2.48 (0.87) | 2.71 (0.78)
  Week 4: Scaling (Head\Neck) (n=352,350,65,66) | 1.43 (1.10) | 1.23 (1.07) | 1.80 (1.16) | 1.94 (1.07)
  Week 4: Scaling (Upper Limbs) (n=352,350,65,66) | 1.88 (0.98) | 1.71 (0.93) | 2.14 (0.68) | 2.42 (0.79)
  Week 4: Scaling (Trunk) (n=352,350,65,66) | 1.79 (1.03) | 1.57 (1.01) | 1.98 (1.01) | 2.41 (0.94)
  Week 4: Scaling (Lower Limbs) (n=352,350,65,66) | 2.11 (0.96) | 1.93 (1.00) | 2.32 (0.92) | 2.64 (0.80)
  Week 8: Erythema (Head\Neck) (n=347,350,65,66) | 1.23 (1.05) | 0.95 (0.98) | 1.92 (1.11) | 1.86 (1.05)
  Week 8: Erythema (Upper Limbs) (n=347,350,65,66) | 1.76 (0.98) | 1.48 (0.93) | 2.43 (0.77) | 2.61 (0.74)
  Week 8: Erythema (Trunk) (n=347,350,65,66) | 1.67 (1.11) | 1.37 (1.02) | 2.31 (1.01) | 2.55 (0.91)
  Week 8: Erythema (Lower Limbs) (n=347,350,65,66) | 1.99 (1.08) | 1.71 (0.98) | 2.62 (0.78) | 2.91 (0.76)
  Week 8: Induration (Head\Neck) (n=347,350,65,66) | 1.04 (1.01) | 0.75 (0.88) | 1.68 (1.03) | 1.67 (1.00)
  Week 8: Induration (Upper Limbs) (n=347,350,65,66) | 1.62 (0.93) | 1.39 (0.93) | 2.15 (0.80) | 2.44 (0.70)
  Week 8: Induration (Trunk) (n=347,350,65,66) | 1.44 (1.02) | 1.26 (1.02) | 2.03 (1.07) | 2.38 (0.99)
  Week 8: Induration (Lower Limbs) (n=347,350,65,66) | 1.74 (1.02) | 1.47 (0.97) | 2.35 (0.87) | 2.67 (0.83)
  Week 8: Scaling (Head\Neck) (n=347,350,65,66) | 1.18 (1.12) | 0.83 (0.97) | 1.80 (1.11) | 1.88 (1.09)
  Week 8: Scaling (Upper Limbs) (n=347,350,65,66) | 1.66 (1.02) | 1.37 (0.96) | 2.05 (0.78) | 2.35 (0.79)
  Week 8: Scaling (Trunk) (n=347,350,65,66) | 1.41 (1.09) | 1.19 (1.05) | 1.83 (1.01) | 2.20 (1.06)
  Week 8: Scaling (Lower Limbs) (n=347,350,65,66) | 1.80 (1.07) | 1.45 (1.03) | 2.22 (0.96) | 2.55 (0.91)
  Week 12: Erythema (Head\Neck) (n=345,345,65,66) | 1.10 (1.09) | 0.83 (0.96) | 1.78 (0.96) | 1.85 (1.00)
  Week 12: Erythema (Upper Limbs) (n=345,345,65,66) | 1.60 (1.07) | 1.28 (0.96) | 2.35 (0.76) | 2.53 (0.75)
  Week 12: Erythema (Trunk) (n=345,345,65,66) | 1.53 (1.18) | 1.12 (1.07) | 2.35 (0.98) | 2.53 (0.95)
  Week 12: Erythema (Lower Limbs) (n=345,345,65,66) | 1.81 (1.13) | 1.39 (1.06) | 2.54 (0.79) | 2.77 (0.86)
  Week 12: Induration (Head\Neck) (n=345,345,65,66) | 0.90 (1.02) | 0.65 (0.86) | 1.54 (0.97) | 1.56 (1.01)
  Week 12: Induration (Upper Limbs)(n=345,345,65,66) | 1.48 (1.02) | 1.17 (0.95) | 2.05 (0.78) | 2.32 (0.84)
  Week 12: Induration (Trunk) (n=345,345,65,66) | 1.34 (1.09) | 0.98 (1.03) | 1.89 (0.99) | 2.27 (0.99)
  Week 12: Induration (Lower Limbs)(n=345,345,65,66) | 1.58 (1.08) | 1.17 (0.98) | 2.26 (0.82) | 2.55 (0.88)
  Week 12: Scaling (Head\Neck) (n=345,345,65,66) | 1.03 (1.06) | 0.72 (0.91) | 1.77 (1.01) | 1.76 (1.10)
  Week 12: Scaling (Upper Limbs) (n=345,345,65,66) | 1.50 (1.07) | 1.18 (0.98) | 2.03 (0.90) | 2.27 (0.83)
  Week 12: Scaling (Trunk) (n=345,345,65,66) | 1.30 (1.12) | 0.95 (1.01) | 1.89 (1.05) | 2.26 (1.09)
  Week 12: Scaling (Lower Limbs) (n=345,345,65,66) | 1.56 (1.10) | 1.14 (0.98) | 2.14 (0.95) | 2.53 (1.00)
  Week 16: Erythema (Head\Neck) (n=323,335,66,66) | 1.01 (1.07) | 0.75 (0.95) | 1.73 (1.05) | 1.91 (1.09)
  Week 16: Erythema (Upper Limbs) (n=323,335,66,66) | 1.46 (1.12) | 1.13 (1.00) | 2.30 (0.80) | 2.53 (0.83)
  Week 16: Erythema (Trunk) (n=323,335,66,66) | 1.40 (1.17) | 1.01 (1.09) | 2.14 (1.11) | 2.58 (1.08)
  Week 16: Erythema (Lower Limbs) (n=323,335,66,66) | 1.63 (1.19) | 1.25 (1.10) | 2.52 (0.83) | 2.82 (0.89)
  Week 16: Induration (Head\Neck) (n=323,335,66,66) | 0.83 (0.97) | 0.60 (0.88) | 1.42 (1.01) | 1.58 (1.12)
  Week 16: Induration (Upper Limbs)(n=323,335,66,66) | 1.34 (1.10) | 1.06 (0.99) | 2.06 (0.87) | 2.33 (0.93)
  Week 16: Induration (Trunk) (n=323,335,66,66) | 1.22 (1.08) | 0.85 (1.05) | 1.83 (1.14) | 2.29 (1.08)
  Week 16: Induration (Lower Limbs)(n=323,335,66,66) | 1.38 (1.07) | 1.01 (1.02) | 2.20 (0.92) | 2.52 (0.86)
  Week 16: Scaling (Head\Neck) (n=323,335,66,66) | 0.94 (1.04) | 0.67 (0.91) | 1.59 (1.02) | 1.76 (1.10)
  Week 16: Scaling (Upper Limbs) (n=323,335,66,66) | 1.41 (1.09) | 1.07 (0.98) | 2.08 (0.90) | 2.29 (0.89)
  Week 16: Scaling (Trunk) (n=323,335,66,66) | 1.15 (1.01) | 0.84 (0.99) | 1.83 (1.12) | 2.12 (1.10)
  Week 16: Scaling (Lower Limbs) (n=323,335,66,66) | 1.42 (1.06) | 1.01 (1.02) | 2.15 (1.00) | 2.50 (1.06)
  Week 20: Erythema (Head\Neck) (n=312,321,66,65) | 0.94 (1.02) | 0.66 (0.94) | 1.08 (0.93) | 1.23 (0.95)
  Week 20: Erythema (Upper Limbs) (n=312,321,66,65) | 1.29 (1.04) | 1.05 (1.01) | 1.48 (0.79) | 1.80 (0.85)
  Week 20: Erythema (Trunk) (n=312,321,66,65) | 1.23 (1.09) | 0.89 (1.06) | 1.36 (0.97) | 1.68 (1.02)
  Week 20: Erythema (Lower Limbs) (n=312,321,66,65) | 1.45 (1.17) | 1.13 (1.09) | 1.71 (0.82) | 1.94 (0.98)
  Week 20: Induration (Head\Neck) (n=312,321,66,65) | 0.78 (0.93) | 0.55 (0.83) | 0.83 (0.83) | 0.97 (0.85)
  Week 20: Induration (Upper Limbs)(n=312,321,66,65) | 1.21 (1.03) | 0.99 (1.00) | 1.38 (0.78) | 1.52 (0.83)
  Week 20: Induration (Trunk) (n=312,321,66,65) | 1.06 (1.03) | 0.78 (1.02) | 1.17 (1.02) | 1.43 (1.02)
  Week 20: Induration (Lower Limbs)(n=312,321,66,65) | 1.24 (1.04) | 0.96 (1.03) | 1.52 (0.85) | 1.66 (1.00)
  Week 20: Scaling (Head\Neck) (n=312,321,66,65) | 0.86 (0.97) | 0.63 (0.94) | 0.98 (0.90) | 1.09 (1.06)
  Week 20: Scaling (Upper Limbs) (n=312,321,66,65) | 1.23 (1.00) | 1.02 (1.03) | 1.50 (0.88) | 1.63 (0.94)
  Week 20: Scaling (Trunk) (n=312,321,66,65) | 0.99 (0.94) | 0.76 (1.00) | 1.20 (1.03) | 1.49 (1.17)
  Week 20: Scaling (Lower Limbs) (n=312,321,66,65) | 1.30 (1.04) | 0.96 (1.03) | 1.55 (1.00) | 1.80 (1.18)
  Week 28: Erythema (Head\Neck) (n=300,307,61,61) | 0.83 (0.99) | 0.65 (0.93) | 0.54 (0.81) | 0.51 (0.87)
  Week 28: Erythema (Upper Limbs) (n=300,307,61,61) | 1.20 (1.08) | 0.96 (1.00) | 1.16 (0.92) | 1.05 (0.88)
  Week 28: Erythema (Trunk) (n=300,307,61,61) | 1.09 (1.14) | 0.77 (1.04) | 0.92 (0.90) | 0.95 (0.97)
  Week 28: Erythema (Lower Limbs) (n=300,307,61,61) | 1.27 (1.19) | 0.97 (1.09) | 1.21 (0.97) | 1.15 (1.00)
  Week 28: Induration (Head\Neck) (n=300,307,61,61) | 0.66 (0.89) | 0.47 (0.76) | 0.44 (0.70) | 0.31 (0.72)
  Week 28: Induration (Upper Limbs)(n=300,307,61,61) | 1.10 (1.05) | 0.90 (1.01) | 1.00 (0.84) | 0.79 (0.82)
  Week 28: Induration (Trunk) (n=300,307,61,61) | 0.93 (1.03) | 0.69 (1.00) | 0.75 (0.85) | 0.80 (1.08)
  Week 28: Induration (Lower Limbs)(n=300,307,61,61) | 1.09 (1.08) | 0.79 (0.99) | 0.98 (0.83) | 0.87 (0.90)
  Week 28: Scaling (Head\Neck) (n=300,307,61,61) | 0.77 (0.95) | 0.57 (0.85) | 0.56 (0.76) | 0.44 (0.85)
  Week 28: Scaling (Upper Limbs) (n=300,307,61,61) | 1.15 (1.06) | 0.90 (0.99) | 1.08 (0.86) | 0.98 (0.92)
  Week 28: Scaling (Trunk) (n=300,307,61,61) | 0.89 (0.97) | 0.64 (0.90) | 0.80 (0.87) | 0.90 (1.14)
  Week 28: Scaling (Lower Limbs) (n=300,307,61,61) | 1.15 (1.07) | 0.79 (0.99) | 1.02 (0.90) | 1.08 (1.08)
  Week 40: Erythema (Head\Neck) (n=203,242,53,47) | 0.55 (0.87) | 0.54 (0.85) | 0.51 (0.87) | 0.32 (0.69)
  Week 40: Erythema (Upper Limbs) (n=203,242,53,47) | 0.87 (0.97) | 0.76 (0.92) | 1.06 (0.93) | 0.55 (0.90)
  Week 40: Erythema (Trunk) (n=203,242,53,47) | 0.68 (0.95) | 0.52 (0.87) | 0.68 (0.89) | 0.57 (0.77)
  Week 40: Erythema (Lower Limbs) (n=203,242,53,47) | 0.88 (1.05) | 0.72 (0.97) | 0.92 (1.00) | 0.55 (0.83)
  Week 40: Induration (Head\Neck) (n=203,242,53,47) | 0.44 (0.73) | 0.45 (0.76) | 0.43 (0.82) | 0.23 (0.52)
  Week 40: Induration (Upper Limbs)(n=203,242,53,47) | 0.79 (0.93) | 0.72 (0.87) | 1.00 (0.88) | 0.36 (0.67)
  Week 40: Induration (Trunk) (n=203,242,53,47) | 0.56 (0.80) | 0.48 (0.81) | 0.57 (0.75) | 0.32 (0.59)
  Week 40: Induration (Lower Limbs)(n=203,242,53,47) | 0.70 (0.91) | 0.62 (0.91) | 0.85 (0.77) | 0.32 (0.59)
  Week 40: Scaling (Head\Neck) (n=203,242,53,47) | 0.53 (0.82) | 0.52 (0.90) | 0.51 (0.78) | 0.30 (0.59)
  Week 40: Scaling (Upper Limbs) (n=203,242,53,47) | 0.85 (0.97) | 0.71 (0.91) | 1.06 (0.82) | 0.49 (0.80)
  Week 40: Scaling (Trunk) (n=203,242,53,47) | 0.53 (0.79) | 0.44 (0.77) | 0.58 (0.75) | 0.47 (0.78)
  Week 40: Scaling (Lower Limbs) (n=203,242,53,47) | 0.78 (0.97) | 0.62 (0.90) | 0.85 (0.86) | 0.45 (0.75)
  Week 52: Erythema (Head\Neck) (n=180,219,47,46) | 0.50 (0.76) | 0.42 (0.78) | 0.55 (0.83) | 0.39 (0.74)
  Week 52: Erythema (Upper Limbs) (n=180,219,47,46) | 0.93 (0.95) | 0.72 (0.87) | 1.06 (0.94) | 0.50 (0.81)
  Week 52: Erythema (Trunk) (n=180,219,47,46) | 0.64 (0.91) | 0.59 (0.93) | 0.66 (0.94) | 0.50 (0.86)
  Week 52: Erythema (Lower Limbs) (n=180,219,47,46) | 0.93 (1.05) | 0.67 (0.98) | 0.87 (0.99) | 0.63 (0.85)
  Week 52: Induration (Head\Neck) (n=180,219,47,46) | 0.47 (0.71) | 0.32 (0.66) | 0.40 (0.68) | 0.24 (0.57)
  Week 52: Induration (Upper Limbs)(n=180,219,47,46) | 0.86 (0.94) | 0.70 (0.87) | 0.98 (0.82) | 0.43 (0.75)
  Week 52: Induration (Trunk) (n=180,219,47,46) | 0.56 (0.81) | 0.54 (0.86) | 0.53 (0.80) | 0.35 (0.77)
  Week 52: Induration (Lower Limbs)(n=180,219,47,46) | 0.84 (0.96) | 0.61 (0.89) | 0.79 (0.88) | 0.39 (0.65)
  Week 52: Scaling (Head\Neck) (n=180,219,47,46) | 0.51 (0.77) | 0.42 (0.78) | 0.62 (0.87) | 0.39 (0.74)
  Week 52: Scaling (Upper Limbs) (n=180,219,47,46) | 0.91 (0.97) | 0.74 (0.88) | 1.06 (0.87) | 0.57 (0.83)
  Week 52: Scaling (Trunk) (n=180,219,47,46) | 0.54 (0.81) | 0.51 (0.79) | 0.57 (0.83) | 0.43 (0.81)
  Week 52: Scaling (Lower Limbs) (n=180,219,47,46) | 0.89 (0.98) | 0.58 (0.90) | 0.91 (0.95) | 0.50 (0.75)

22. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Component Scores at Week 2, 4, 8, 12, 16, 20, 28, 40 and 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. Basic characteristics of psoriatic lesions: erythema, induration, and scaling (PASI components) are scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]) according to a 5-point scale: 0 (no involvement); 1 (slight); 2 (moderate); 3 (marked); 4 (very marked). PASI component score range from 0 to 4, where higher scores indicate greater severity of psoriatic lesions.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
units on a scale
  Week 2: Erythema (Head\Neck) (n=358,358,66,64) | -0.45 (0.78) | -0.51 (0.82) | -0.24 (0.61) | -0.06 (0.66)
  Week 2: Erythema (Upper Limbs) (n=358,358,66,64) | -0.46 (0.68) | -0.63 (0.71) | -0.20 (0.47) | -0.09 (0.56)
  Week 2: Erythema (Trunk) (n=358,358,66,64) | -0.46 (0.69) | -0.63 (0.74) | -0.21 (0.51) | -0.17 (0.49)
  Week 2: Erythema (Lower Limbs) (n=358,358,66,64) | -0.47 (0.70) | -0.59 (0.74) | -0.15 (0.44) | -0.13 (0.58)
  Week 2: Induration (Head\Neck) (n=358,358,66,64) | -0.37 (0.67) | -0.48 (0.78) | -0.20 (0.53) | -0.08 (0.57)
  Week 2: Induration (Upper Limbs) (n=358,358,66,64) | -0.42 (0.67) | -0.53 (0.74) | -0.35 (0.62) | -0.11 (0.54)
  Week 2: Induration (Trunk) (n=358,358,66,64) | -0.40 (0.72) | -0.53 (0.74) | -0.21 (0.48) | -0.14 (0.50)
  Week 2: Induration (Lower Limbs) (n=358,358,66,64) | -0.41 (0.66) | -0.52 (0.65) | -0.21 (0.45) | -0.27 (0.48)
  Week 2: Scaling (Head\Neck) (n=358,358,66,64) | -0.47 (0.67) | -0.56 (0.86) | -0.30 (0.80) | -0.17 (0.55)
  Week 2: Scaling (Upper Limbs) (n=358,358,66,64) | -0.45 (0.72) | -0.63 (0.81) | -0.29 (0.55) | -0.20 (0.72)
  Week 2: Scaling (Trunk) (n=358,358,66,64) | -0.48 (0.75) | -0.60 (0.81) | -0.23 (0.70) | -0.30 (0.61)
  Week 2: Scaling (Lower Limbs) (n=358,358,66,64) | -0.48 (0.74) | -0.57 (0.74) | -0.24 (0.66) | -0.23 (0.61)
  Week 4: Erythema (Head\Neck) (n=352,350,65,66) | -0.84 (1.04) | -0.90 (1.01) | -0.48 (0.87) | -0.33 (0.71)
  Week 4: Erythema (Upper Limbs) (n=352,350,65,66) | -0.86 (0.88) | -1.03 (0.84) | -0.42 (0.73) | -0.20 (0.64)
  Week 4: Erythema (Trunk) (n=352,350,65,66) | -0.86 (0.88) | -1.08 (0.95) | -0.37 (0.86) | -0.33 (0.59)
  Week 4: Erythema (Lower Limbs) (n=352,350,65,66) | -0.86 (0.89) | -1.04 (0.87) | -0.35 (0.62) | -0.30 (0.70)
  Week 4: Induration (Head\Neck) (n=352,350,65,66) | -0.79 (0.97) | -0.85 (1.00) | -0.40 (0.68) | -0.27 (0.69)
  Week 4: Induration (Upper Limbs) (n=352,350,65,66) | -0.82 (0.88) | -0.91 (0.85) | -0.46 (0.69) | -0.15 (0.66)
  Week 4: Induration (Trunk) (n=352,350,65,66) | -0.79 (0.89) | -0.95 (0.90) | -0.37 (0.88) | -0.18 (0.63)
  Week 4: Induration (Lower Limbs) (n=352,350,65,66) | -0.85 (0.85) | -0.96 (0.82) | -0.35 (0.60) | -0.27 (0.62)
  Week 4: Scaling (Head\Neck) (n=352,350,65,66) | -0.88 (1.00) | -0.99 (1.07) | -0.54 (0.95) | -0.30 (0.74)
  Week 4: Scaling (Upper Limbs) (n=352,350,65,66) | -0.86 (0.97) | -1.00 (0.93) | -0.40 (0.72) | -0.33 (0.73)
  Week 4: Scaling (Trunk) (n=352,350,65,66) | -0.81 (0.93) | -1.03 (0.96) | -0.37 (0.84) | -0.36 (0.69)
  Week 4: Scaling (Lower Limbs) (n=352,350,65,66) | -0.87 (0.96) | -0.97 (0.94) | -0.45 (0.73) | -0.33 (0.71)
  Week 8: Erythema (Head\Neck) (n=347,350,65,66) | -1.05 (1.16) | -1.28 (1.11) | -0.45 (1.03) | -0.39 (0.99)
  Week 8: Erythema (Upper Limbs) (n=347,350,65,66) | -1.10 (1.04) | -1.41 (0.99) | -0.40 (0.70) | -0.32 (0.73)
  Week 8: Erythema (Trunk) (n=347,350,65,66) | -1.18 (1.10) | -1.54 (1.03) | -0.52 (0.87) | -0.53 (0.81)
  Week 8: Erythema (Lower Limbs) (n=347,350,65,66) | -1.22 (1.10) | -1.48 (1.00) | -0.51 (0.73) | -0.36 (0.65)
  Week 8: Induration (Head\Neck) (n=347,350,65,66) | -1.02 (1.10) | -1.21 (1.10) | -0.45 (0.87) | -0.35 (1.03)
  Week 8: Induration (Upper Limbs) (n=347,350,65,66) | -1.07 (0.98) | -1.26 (0.99) | -0.55 (0.75) | -0.24 (0.66)
  Week 8: Induration (Trunk) (n=347,350,65,66) | -1.14 (1.05) | -1.36 (1.06) | -0.54 (0.89) | -0.33 (0.88)
  Week 8: Induration (Lower Limbs) (n=347,350,65,66) | -1.16 (1.06) | -1.42 (0.99) | -0.48 (0.69) | -0.32 (0.79)
  Week 8: Scaling (Head\Neck) (n=347,350,65,66) | -1.12 (1.17) | -1.39 (1.16) | -0.52 (1.03) | -0.36 (1.06)
  Week 8: Scaling (Upper Limbs) (n=347,350,65,66) | -1.08 (1.07) | -1.33 (1.08) | -0.49 (0.77) | -0.41 (0.86)
  Week 8: Scaling (Trunk) (n=347,350,65,66) | -1.18 (1.11) | -1.40 (1.12) | -0.57 (0.87) | -0.58 (0.86)
  Week 8: Scaling (Lower Limbs) (n=347,350,65,66) | -1.17 (1.11) | -1.44 (1.09) | -0.55 (0.81) | -0.42 (0.84)
  Week 12: Erythema (Head\Neck) (n=345,345,65,66) | -1.18 (1.21) | -1.41 (1.16) | -0.58 (1.03) | -0.41 (0.96)
  Week 12: Erythema (Upper Limbs) (n=345,345,65,66) | -1.26 (1.15) | -1.61 (1.06) | -0.48 (0.79) | -0.39 (0.72)
  Week 12: Erythema (Trunk) (n=345,345,65,66) | -1.32 (1.22) | -1.80 (1.15) | -0.43 (1.00) | -0.55 (0.83)
  Week 12: Erythema (Lower Limbs) (n=345,345,65,66) | -1.40 (1.17) | -1.79 (1.10) | -0.60 (0.72) | -0.50 (0.79)
  Week 12: Induration (Head\Neck) (n=345,345,65,66) | -1.16 (1.18) | -1.32 (1.15) | -0.60 (0.97) | -0.45 (0.91)
  Week 12: Induration (Upper Limbs)(n=345,345,65,66) | -1.21 (1.14) | -1.47 (1.05) | -0.66 (0.78) | -0.36 (0.82)
  Week 12: Induration (Trunk) (n=345,345,65,66) | -1.25 (1.17) | -1.65 (1.14) | -0.63 (0.88) | -0.44 (0.90)
  Week 12: Induration (Lower Limbs)(n=345,345,65,66) | -1.33 (1.18) | -1.72 (1.09) | -0.57 (0.68) | -0.44 (0.84)
  Week 12: Scaling (Head\Neck) (n=345,345,65,66) | -1.28 (1.20) | -1.52 (1.20) | -0.57 (1.06) | -0.48 (1.08)
  Week 12: Scaling (Upper Limbs) (n=345,345,65,66) | -1.24 (1.22) | -1.52 (1.17) | -0.51 (0.95) | -0.48 (0.83)
  Week 12: Scaling (Trunk) (n=345,345,65,66) | -1.30 (1.19) | -1.65 (1.16) | -0.46 (0.90) | -0.52 (0.88)
  Week 12: Scaling (Lower Limbs) (n=345,345,65,66) | -1.41 (1.17) | -1.76 (1.13) | -0.63 (0.84) | -0.44 (0.95)
  Week 16: Erythema (Head\Neck) (n=323,335,66,66) | -1.28 (1.26) | -1.48 (1.19) | -0.65 (0.97) | -0.35 (1.02)
  Week 16: Erythema (Upper Limbs) (n=323,335,66,66) | -1.41 (1.19) | -1.76 (1.12) | -0.53 (0.86) | -0.39 (0.74)
  Week 16: Erythema (Trunk) (n=323,335,66,66) | -1.45 (1.23) | -1.90 (1.18) | -0.65 (1.10) | -0.50 (1.00)
  Week 16: Erythema (Lower Limbs) (n=323,335,66,66) | -1.59 (1.23) | -1.94 (1.17) | -0.62 (0.84) | -0.45 (0.79)
  Week 16: Induration (Head\Neck) (n=323,335,66,66) | -1.22 (1.22) | -1.37 (1.16) | -0.71 (1.00) | -0.44 (1.10)
  Week 16: Induration (Upper Limbs)(n=323,335,66,66) | -1.35 (1.19) | -1.58 (1.14) | -0.65 (0.83) | -0.35 (0.95)
  Week 16: Induration (Trunk) (n=323,335,66,66) | -1.37 (1.18) | -1.75 (1.21) | -0.70 (1.01) | -0.42 (0.95)
  Week 16: Induration (Lower Limbs)(n=323,335,66,66) | -1.54 (1.22) | -1.88 (1.19) | -0.64 (0.76) | -0.47 (0.92)
  Week 16: Scaling (Head\Neck) (n=323,335,66,66) | -1.37 (1.26) | -1.57 (1.24) | -0.74 (1.06) | -0.48 (1.01)
  Week 16: Scaling (Upper Limbs) (n=323,335,66,66) | -1.35 (1.22) | -1.63 (1.20) | -0.47 (0.88) | -0.47 (0.88)
  Week 16: Scaling (Trunk) (n=323,335,66,66) | -1.44 (1.16) | -1.76 (1.17) | -0.53 (1.00) | -0.65 (0.89)
  Week 16: Scaling (Lower Limbs) (n=323,335,66,66) | -1.56 (1.17) | -1.89 (1.22) | -0.62 (0.91) | -0.47 (1.01)
  Week 20: Erythema (Head\Neck) (n=312,321,66,65) | -1.37 (1.20) | -1.57 (1.25) | -1.30 (0.99) | -1.02 (0.99)
  Week 20: Erythema (Upper Limbs) (n=312,321,66,65) | -1.58 (1.18) | -1.84 (1.13) | -1.35 (0.92) | -1.12 (0.93)
  Week 20: Erythema (Trunk) (n=312,321,66,65) | -1.63 (1.20) | -2.03 (1.16) | -1.42 (1.02) | -1.40 (1.06)
  Week 20: Erythema (Lower Limbs) (n=312,321,66,65) | -1.77 (1.20) | -2.06 (1.18) | -1.42 (0.82) | -1.34 (1.08)
  Week 20: Induration (Head\Neck) (n=312,321,66,65) | -1.29 (1.20) | -1.44 (1.18) | -1.30 (0.96) | -1.03 (1.03)
  Week 20: Induration (Upper Limbs)(n=312,321,66,65) | -1.48 (1.18) | -1.65 (1.13) | -1.33 (0.79) | -1.15 (1.00)
  Week 20: Induration (Trunk) (n=312,321,66,65) | -1.53 (1.16) | -1.83 (1.21) | -1.36 (1.00) | -1.28 (0.96)
  Week 20: Induration (Lower Limbs)(n=312,321,66,65) | -1.68 (1.22) | -1.93 (1.21) | -1.32 (0.95) | -1.32 (1.05)
  Week 20: Scaling (Head\Neck) (n=312,321,66,65) | -1.47 (1.21) | -1.63 (1.26) | -1.35 (1.17) | -1.15 (1.11)
  Week 20: Scaling (Upper Limbs) (n=312,321,66,65) | -1.52 (1.18) | -1.69 (1.21) | -1.05 (1.01) | -1.14 (1.13)
  Week 20: Scaling (Trunk) (n=312,321,66,65) | -1.60 (1.12) | -1.84 (1.20) | -1.17 (1.02) | -1.28 (1.10)
  Week 20: Scaling (Lower Limbs) (n=312,321,66,65) | -1.68 (1.19) | -1.94 (1.23) | -1.23 (1.11) | -1.18 (1.16)
  Week 28: Erythema (Head\Neck) (n=300,307,61,61) | -1.47 (1.24) | -1.59 (1.23) | -1.80 (1.08) | -1.70 (0.99)
  Week 28: Erythema (Upper Limbs) (n=300,307,61,61) | -1.67 (1.24) | -1.92 (1.13) | -1.67 (1.04) | -1.89 (1.00)
  Week 28: Erythema (Trunk) (n=300,307,61,61) | -1.77 (1.29) | -2.15 (1.17) | -1.89 (0.98) | -2.13 (1.02)
  Week 28: Erythema (Lower Limbs) (n=300,307,61,61) | -1.95 (1.22) | -2.23 (1.22) | -1.92 (0.99) | -2.11 (0.98)
  Week 28: Induration (Head\Neck) (n=300,307,61,61) | -1.40 (1.20) | -1.53 (1.16) | -1.69 (1.13) | -1.64 (1.03)
  Week 28: Induration (Upper Limbs)(n=300,307,61,61) | -1.58 (1.23) | -1.75 (1.13) | -1.70 (0.95) | -1.92 (1.02)
  Week 28: Induration (Trunk) (n=300,307,61,61) | -1.66 (1.19) | -1.92 (1.21) | -1.80 (1.01) | -1.93 (1.14)
  Week 28: Induration (Lower Limbs)(n=300,307,61,61) | -1.81 (1.27) | -2.11 (1.21) | -1.89 (1.00) | -2.11 (1.10)
  Week 28: Scaling (Head\Neck) (n=300,307,61,61) | -1.55 (1.28) | -1.71 (1.23) | -1.72 (1.29) | -1.79 (1.13)
  Week 28: Scaling (Upper Limbs) (n=300,307,61,61) | -1.59 (1.28) | -1.81 (1.22) | -1.48 (1.03) | -1.84 (1.07)
  Week 28: Scaling (Trunk) (n=300,307,61,61) | -1.72 (1.23) | -1.97 (1.14) | -1.61 (1.07) | -1.90 (1.14)
  Week 28: Scaling (Lower Limbs) (n=300,307,61,61) | -1.81 (1.24) | -2.12 (1.21) | -1.80 (1.09) | -1.95 (1.12)
  Week 40: Erythema (Head\Neck) (n=203,242,53,47) | -1.78 (1.15) | -1.69 (1.16) | -1.83 (1.14) | -1.81 (1.15)
  Week 40: Erythema (Upper Limbs) (n=203,242,53,47) | -2.02 (1.15) | -2.11 (1.09) | -1.75 (1.12) | -2.40 (0.99)
  Week 40: Erythema (Trunk) (n=203,242,53,47) | -2.19 (1.14) | -2.40 (1.03) | -2.11 (0.95) | -2.45 (0.93)
  Week 40: Erythema (Lower Limbs) (n=203,242,53,47) | -2.34 (1.10) | -2.45 (1.11) | -2.21 (1.10) | -2.68 (0.89)
  Week 40: Induration (Head\Neck) (n=203,242,53,47) | -1.68 (1.10) | -1.56 (1.14) | -1.72 (1.26) | -1.72 (1.16)
  Week 40: Induration (Upper Limbs)(n=203,242,53,47) | -1.94 (1.09) | -1.93 (1.04) | -1.70 (1.01) | -2.32 (0.98)
  Week 40: Induration (Trunk) (n=203,242,53,47) | -2.09 (1.02) | -2.15 (1.10) | -2.00 (0.98) | -2.30 (1.10)
  Week 40: Induration (Lower Limbs)(n=203,242,53,47) | -2.29 (1.10) | -2.28 (1.15) | -2.04 (1.00) | -2.64 (1.03)
  Week 40: Scaling (Head\Neck) (n=203,242,53,47) | -1.85 (1.18) | -1.77 (1.27) | -1.87 (1.35) | -1.96 (1.23)
  Week 40: Scaling (Upper Limbs) (n=203,242,53,47) | -1.95 (1.22) | -2.01 (1.19) | -1.55 (0.99) | -2.34 (1.05)
  Week 40: Scaling (Trunk) (n=203,242,53,47) | -2.15 (1.07) | -2.20 (1.07) | -1.81 (1.06) | -2.26 (1.01)
  Week 40: Scaling (Lower Limbs) (n=203,242,53,47) | -2.20 (1.16) | -2.30 (1.19) | -2.00 (1.09) | -2.57 (0.90)
  Week 52: Erythema (Head\Neck) (n=180,219,47,46) | -1.81 (1.08) | -1.75 (1.18) | -1.70 (1.20) | -1.74 (1.04)
  Week 52: Erythema (Upper Limbs) (n=180,219,47,46) | -1.95 (1.13) | -2.13 (1.04) | -1.77 (1.16) | -2.46 (0.98)
  Week 52: Erythema (Trunk) (n=180,219,47,46) | -2.22 (1.12) | -2.31 (1.13) | -2.15 (1.02) | -2.52 (1.03)
  Week 52: Erythema (Lower Limbs) (n=180,219,47,46) | -2.29 (1.16) | -2.50 (1.12) | -2.26 (1.13) | -2.61 (0.98)
  Week 52: Induration (Head\Neck) (n=180,219,47,46) | -1.65 (1.11) | -1.69 (1.13) | -1.68 (1.09) | -1.72 (1.13)
  Week 52: Induration (Upper Limbs)(n=180,219,47,46) | -1.86 (1.12) | -1.95 (1.07) | -1.70 (1.04) | -2.24 (1.02)
  Week 52: Induration (Trunk) (n=180,219,47,46) | -2.08 (1.03) | -2.11 (1.16) | -2.04 (1.04) | -2.24 (1.14)
  Week 52: Induration (Lower Limbs)(n=180,219,47,46) | -2.17 (1.17) | -2.30 (1.18) | -2.13 (1.10) | -2.54 (1.03)
  Week 52: Scaling (Head\Neck) (n=180,219,47,46) | -1.86 (1.16) | -1.87 (1.23) | -1.68 (1.29) | -1.89 (1.20)
  Week 52: Scaling (Upper Limbs) (n=180,219,47,46) | -1.87 (1.20) | -1.99 (1.11) | -1.53 (1.10) | -2.26 (1.00)
  Week 52: Scaling (Trunk) (n=180,219,47,46) | -2.17 (1.05) | -2.16 (1.08) | -1.85 (1.12) | -2.28 (1.07)
  Week 52: Scaling (Lower Limbs) (n=180,219,47,46) | -2.12 (1.16) | -2.35 (1.16) | -1.98 (1.24) | -2.52 (0.98)

23. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 2, 4, 8, 12, 16, 20, 28, 40 and 52
Description: as for outcome 19
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 359 | 358 | 66 | 66
percent change
  Change at Week 2 | -18.50 (1.11) | -24.86 (1.11) | -8.99 (2.59) | -5.85 (2.61)
  Change at Week 4 | -34.60 (1.45) | -43.08 (1.46) | -15.75 (3.38) | -10.76 (3.38)
  Change at Week 8 | -47.72 (1.68) | -60.48 (1.68) | -20.27 (3.89) | -13.02 (3.88)
  Change at Week 12 | -54.07 (1.83) | -69.11 (1.83) | -23.02 (4.21) | -15.26 (4.21)
  Change at Week 16 | -57.25 (1.97) | -72.71 (1.96) | -25.66 (4.51) | -13.33 (4.51)
  Change at Week 20 | -63.73 (1.74) | -75.05 (1.73) | -56.71 (3.93) | -49.48 (3.94)
  Change at Week 28 | -68.62 (1.69) | -78.91 (1.67) | -73.49 (3.75) | -76.64 (3.78)
  Change at Week 40 | -67.06 (1.82) | -76.36 (1.77) | -73.52 (3.93) | -81.21 (4.01)
  Change at Week 52 | -64.15 (1.91) | -74.61 (1.85) | -70.60 (4.11) | -80.94 (4.17)

24. Secondary Outcome: Total Body Surface Area (BSA) With Psoriasis
Description: as for outcome 3
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
percentage of BSA
  Baseline (n = 363, 360, 66, 66) | 28.48 (16.42) | 31.13 (17.64) | 28.03 (16.99) | 30.17 (16.34)
  Week 2 (n = 358, 358, 66, 64) | 27.08 (16.85) | 27.86 (17.24) | 28.21 (19.27) | 30.32 (16.99)
  Week 4 (n = 352, 350, 65, 66) | 23.69 (16.56) | 22.79 (17.52) | 27.15 (20.08) | 29.52 (17.01)
  Week 8 (n = 347, 350, 65, 66) | 18.99 (16.28) | 16.49 (16.23) | 26.82 (19.93) | 29.43 (17.45)
  Week 12 (n = 345, 345, 65, 66) | 15.73 (16.03) | 12.64 (15.01) | 25.89 (20.50) | 29.02 (17.58)
  Week 16 (n = 323, 335, 66, 66) | 13.08 (15.75) | 9.48 (12.99) | 25.89 (21.77) | 29.14 (19.18)
  Week 20 (n = 312, 321, 66, 65) | 10.77 (14.23) | 7.59 (11.45) | 18.57 (20.49) | 21.73 (17.48)
  Week 28 (n = 300, 307, 61, 61) | 8.92 (13.07) | 6.05 (9.36) | 9.54 (15.85) | 9.96 (12.39)
  Week 40 (n = 203, 242, 53, 47) | 4.37 (7.58) | 3.51 (6.03) | 4.47 (6.96) | 3.02 (4.19)
  Week 52 (n = 180, 219, 47, 46) | 4.42 (6.93) | 2.94 (5.29) | 3.79 (4.37) | 2.09 (2.80)

25. Secondary Outcome: Percent Change From Baseline in Total Body Surface Area (BSA) With Psoriasis at Week 2, 4, 8, 12, 16, 20, 28, 40 and 52
Description: as for outcome 3
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 359 | 358 | 66 | 66
percent change
  Change at Week 2 | -6.89 (0.97) | -10.44 (0.97) | -1.92 (2.25) | -1.23 (2.27)
  Change at Week 4 | -18.31 (1.58) | -26.73 (1.58) | -5.29 (3.67) | -1.81 (3.66)
  Change at Week 8 | -34.86 (1.93) | -46.27 (1.93) | -6.73 (4.46) | -1.57 (4.45)
  Change at Week 12 | -45.72 (2.13) | -59.20 (2.13) | -9.62 (4.91) | -0.84 (4.91)
  Change at Week 16 | -51.87 (2.41) | -67.12 (2.41) | -11.22 (5.50) | 2.03 (5.50)
  Change at Week 20 | -58.67 (2.22) | -71.96 (2.21) | -37.66 (5.03) | -26.49 (5.04)
  Change at Week 28 | -64.74 (2.27) | -76.82 (2.24) | -66.75 (5.03) | -64.11 (5.07)
  Change at Week 40 | -73.29 (1.72) | -80.78 (1.67) | -73.67 (3.69) | -79.92 (3.78)
  Change at Week 52 | -74.95 (1.55) | -82.36 (1.48) | -74.84 (3.26) | -84.79 (3.33)

26. Secondary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 50 (PASI 50) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 50 response was defined as at least 50% reduction in PASI relative to Baseline. Percentage of participants with PASI 50 response is reported.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
percentage of participants
  Week 2 | 9.09 [6.13 to 12.05] | 17.22 [13.32 to 21.12] | 3.03 [0.00 to 7.17] | 0.00 [0.00 to 0.00]
  Week 4 | 28.65 [24.00 to 33.30] | 39.72 [34.67 to 44.78] | 9.09 [2.16 to 16.03] | 1.52 [0.00 to 4.46]
  Week 8 | 47.93 [42.79 to 53.07] | 65.56 [60.65 to 70.46] | 18.18 [8.88 to 27.49] | 12.12 [4.25 to 20.00]
  Week 12 | 58.95 [53.89 to 64.01] | 73.89 [69.35 to 78.43] | 24.24 [13.90 to 34.58] | 12.12 [4.25 to 20.00]
  Week 16 | 60.33 [55.30 to 65.36] | 76.94 [72.59 to 81.30] | 22.73 [12.62 to 32.84] | 21.21 [11.35 to 31.08]
  Week 20 | 66.12 [61.25 to 70.98] | 75.83 [71.41 to 80.26] | 63.64 [52.03 to 75.24] | 54.55 [42.53 to 66.56]
  Week 28 | 66.39 [61.53 to 71.25] | 76.11 [71.71 to 80.52] | 77.27 [67.16 to 87.38] | 83.33 [74.34 to 92.32]
  Week 40 | 53.99 [48.87 to 59.12] | 63.61 [58.64 to 68.58] | 75.76 [65.42 to 86.10] | 71.21 [60.29 to 82.14]
  Week 52 | 48.21 [43.07 to 53.35] | 59.44 [54.37 to 64.52] | 66.67 [55.29 to 78.04] | 69.70 [58.61 to 80.78]

27. Secondary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 90 (PASI 90) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 90 response was defined as at least 90% reduction in PASI relative to Baseline. Percentage of participants with PASI 90 response up to Week 52 is reported.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
percentage of participants
  Week 2 | 0.28 [0.00 to 0.81] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 4 | 1.65 [0.34 to 2.96] | 3.89 [1.89 to 5.89] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 8 | 9.64 [6.61 to 12.68] | 18.61 [14.59 to 22.63] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 12 | 15.43 [11.71 to 19.14] | 28.06 [23.41 to 32.70] | 1.52 [0.00 to 4.46] | 0.00 [0.00 to 0.00]
  Week 16 | 19.83 [15.73 to 23.94] | 39.44 [34.40 to 44.49] | 0.00 [0.00 to 0.00] | 1.52 [0.00 to 4.46]
  Week 20 | 23.14 [18.80 to 27.48] | 40.28 [35.21 to 45.34] | 7.58 [1.19 to 13.96] | 9.09 [2.16 to 16.03]
  Week 28 | 31.13 [26.37 to 35.89] | 43.61 [38.49 to 48.73] | 25.76 [15.21 to 36.31] | 39.39 [27.61 to 51.18]
  Week 40 | 28.10 [23.48 to 32.72] | 41.39 [36.30 to 46.48] | 34.85 [23.35 to 46.34] | 54.55 [42.53 to 66.56]
  Week 52 | 23.42 [19.06 to 27.77] | 36.94 [31.96 to 41.93] | 31.82 [20.58 to 43.06] | 53.03 [40.99 to 65.07]

28. Secondary Outcome: Percentage of Participants With Psoriasis Area and Severity Index (PASI) Score of at Least 125% of Baseline PASI Score
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. Percentage of participants with PASI score of at least 125% of baseline PASI score are reported.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
percentage of participants
  Week 2 (n = 358, 358, 66, 64) | 0.56 [0.00 to 1.33] | 1.12 [0.03 to 2.21] | 4.55 [0.00 to 9.57] | 3.13 [0.00 to 7.39]
  Week 4 (n = 352, 350, 65, 66) | 1.14 [0.03 to 2.24] | 0.57 [0.00 to 1.36] | 1.54 [0.00 to 4.53] | 4.55 [0.00 to 9.57]
  Week 8 (n = 347, 350, 65, 66) | 2.02 [0.54 to 3.50] | 0.29 [0.00 to 0.84] | 3.08 [0.00 to 7.28] | 7.58 [1.19 to 13.96]
  Week 12 (n = 345, 345, 65, 66) | 2.90 [1.13 to 4.67] | 1.16 [0.03 to 2.29] | 6.15 [0.31 to 12.00] | 9.09 [2.16 to 16.03]
  Week 16 (n = 323, 335, 66, 66) | 2.48 [0.78 to 4.17] | 0.90 [0.00 to 1.90] | 6.06 [0.30 to 11.82] | 12.12 [4.25 to 20.00]
  Week 20 (n = 312, 321, 66, 65) | 1.60 [0.21 to 3.00] | 0.62 [0.00 to 1.48] | 1.52 [0.00 to 4.46] | 4.62 [0.00 to 9.72]
  Week 28 (n = 300, 307, 61, 61) | 1.00 [0.00 to 2.13] | 0.33 [0.00 to 0.96] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 40 (n = 203, 242, 53, 47) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 52 (n = 180, 219, 47, 46) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

29. Secondary Outcome: Nail Psoriasis Severity Index (NAPSI) Score
Description: as for outcome 9
Time Frame: Baseline, Week 8, 16, 20, 28, 40, 52
Population: FAS. Analysis population for "Placebo, CP-690,550" groups included FAS participants who were re-randomized at Week 16 to receive CP-690,550 5 mg or 10 mg. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies participants evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 247 | 250 | 34 | 46
units on a scale
  Baseline (n=247,250,34,46) | 26.64 (20.65) | 28.24 (20.89) | 26.76 (18.33) | 23.91 (16.21)
  Week 8 (n=236,242,33,46) | 24.32 (20.60) | 22.47 (19.43) | 25.55 (18.50) | 24.61 (16.76)
  Week 16 (n=215,233,34,46) | 20.09 (18.79) | 16.53 (17.87) | 27.82 (17.64) | 25.46 (18.57)
  Week 20 (n=210,227,34,45) | 16.53 (17.35) | 12.96 (16.11) | 23.97 (18.18) | 21.18 (18.69)
  Week 28 (n=202,213,30,44) | 13.42 (16.17) | 9.49 (13.92) | 16.77 (14.69) | 14.77 (17.29)
  Week 40 (n=125,167,24,33) | 7.36 (10.04) | 7.19 (12.71) | 5.67 (7.92) | 8.85 (11.27)
  Week 52 (n=110,148,21,32) | 6.94 (9.48) | 6.73 (12.44) | 5.90 (8.92) | 6.66 (9.09)

30. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI) Score at Week 8, 16, 20, 28, 40 and 52
Description: as for outcome 9
Time Frame: Baseline, Week 8, 16, 20, 28, 40, 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 247 | 250 | 34 | 46
units on a scale
  Change at Week 8 (n= 236, 242, 33, 46) | -2.58 (10.98) | -5.55 (12.64) | -0.82 (7.26) | 0.70 (6.89)
  Change at Week 16 (n= 215, 233, 34, 46) | -6.91 (13.93) | -11.70 (16.68) | 1.06 (9.37) | 1.54 (11.34)
  Change at Week 20 (n= 210, 227, 34, 45) | -10.51 (15.17) | -15.16 (17.51) | -2.79 (11.83) | -2.53 (13.00)
  Change at Week 28 (n= 202, 213, 30, 44) | -13.08 (16.53) | -19.07 (18.62) | -10.30 (13.90) | -8.50 (14.18)
  Change at Week 40 (n= 125, 167, 24, 33) | -18.40 (17.47) | -21.63 (19.61) | -16.38 (15.34) | -13.21 (13.07)
  Change at Week 52 (n= 110, 148, 21, 32) | -18.49 (17.03) | -22.28 (20.33) | -17.19 (14.32) | -15.97 (12.47)

31. Secondary Outcome: Number of Affected Nails
Description: Nail psoriasis is evaluated by the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Total number psoriasis affected nails (presence of psoriatic manifestations on the nail matrix/nail bed) were assessed and reported.
Time Frame: Baseline, Week 8, 16, 20, 28, 40, 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: nails
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 247 | 250 | 34 | 46
nails
  Baseline (n= 247, 250, 34, 46) | 7.21 (3.14) | 7.71 (3.12) | 7.73 (3.05) | 7.24 (3.39)
  Week 8 (n= 234, 242, 32, 46) | 6.87 (3.58) | 6.65 (3.80) | 8.00 (3.01) | 7.48 (3.00)
  Week 16 (n= 215, 233, 33, 45) | 6.25 (3.79) | 5.44 (4.16) | 8.27 (2.65) | 7.56 (3.03)
  Week 20 (n= 209, 227, 33, 44) | 5.53 (3.83) | 4.65 (4.13) | 7.48 (3.01) | 6.43 (3.70)
  Week 28 (n= 202, 213, 30, 44) | 4.77 (3.92) | 3.76 (4.03) | 6.63 (3.32) | 5.09 (3.84)
  Week 40 (n= 125, 167, 24, 33) | 3.49 (3.68) | 2.91 (3.61) | 3.13 (3.69) | 3.94 (4.00)
  Week 52 (n= 110, 148, 21, 32) | 3.44 (3.60) | 2.64 (3.57) | 3.10 (3.70) | 3.25 (3.88)

32. Secondary Outcome: Percent Change From Baseline in Nail Psoriasis Severity Index (NAPSI) Score at Week 8, 16, 20, 28, 40 and 52
Description: as for outcome 9
Time Frame: Baseline, Week 8, 16, 20, 28, 40, 52
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 238 | 242 | 34 | 46
percent change
  Percent Change at Week 8 | 2.58 (6.46) | -19.37 (6.40) | 16.91 (17.18) | 36.22 (14.67)
  Percent Change at Week 16 | -14.13 (9.39) | -42.26 (9.16) | 78.80 (24.22) | 50.19 (20.82)
  Percent Change at Week 20 | -32.74 (9.20) | -52.62 (8.93) | 43.82 (23.46) | 38.66 (20.24)
  Percent Change at Week 28 | -43.52 (7.22) | -65.20 (7.06) | 12.39 (18.71) | -18.71 (15.95)
  Percent Change at Week 40 | -64.55 (4.05) | -75.41 (3.57) | -57.01 (9.38) | -54.83 (8.02)
  Percent Change at Week 52 | -58.27 (5.98) | -73.56 (5.54) | -45.67 (14.67) | -72.42 (12.31)

33. Secondary Outcome: Percentage of Participants With Nail Psoriasis Severity Index 75 (NAPSI 75) Response
Description: The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each finger nail divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores = more severe psoriasis. NAPSI 75 response was defined as at least a 75% reduction in NAPSI relative to Baseline. Percentage of participants with NAPSI 75 response is reported.
Time Frame: Week 8, 16, 20, 28, 40, 52
Population: FAS. Analysis population for "Placebo, CP-690,550" groups included FAS participants who were re-randomized at Week 16 to receive CP-690,550 5 mg or 10 mg. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. NRI method was used to impute missing values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 247 | 250 | 34 | 46
percentage of participants
  Week 8 | 9.72 [6.02 to 13.41] | 14.40 [10.05 to 18.75] | 8.82 [0.00 to 18.36] | 4.35 [0.00 to 10.24]
  Week 16 | 14.98 [10.53 to 19.43] | 29.20 [23.56 to 34.84] | 5.88 [0.00 to 13.79] | 6.52 [0.00 to 13.66]
  Week 20 | 21.05 [15.97 to 26.14] | 39.20 [33.15 to 45.25] | 8.82 [0.00 to 18.36] | 23.91 [11.59 to 36.24]
  Week 28 | 31.17 [25.40 to 36.95] | 49.20 [43.00 to 55.40] | 17.65 [4.83 to 30.46] | 28.26 [15.25 to 41.27]
  Week 40 | 28.34 [22.72 to 33.96] | 48.80 [42.60 to 55.00] | 41.18 [24.63 to 57.72] | 36.96 [23.01 to 50.91]
  Week 52 | 25.51 [20.07 to 30.94] | 41.20 [35.10 to 47.30] | 35.29 [19.23 to 51.36] | 43.48 [29.15 to 57.80]

34. Secondary Outcome: Percentage of Participants With Nail Psoriasis Severity Index 100 (NAPSI 100) Response
Description: The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each finger nail divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores = more severe psoriasis. NAPSI 100 response was defined as at least a 100% reduction in NAPSI relative to Baseline. Percentage of participants with NAPSI 100 response is reported.
Time Frame: Week 8, 16, 20, 28, 40, 52
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 247 | 250 | 34 | 46
percentage of participants
  Week 8 | 8.10 [4.70 to 11.50] | 12.40 [8.31 to 16.49] | 5.88 [0.00 to 13.79] | 4.35 [0.00 to 10.24]
  Week 16 | 10.12 [6.36 to 13.88] | 20.00 [15.04 to 24.96] | 5.88 [0.00 to 13.79] | 4.35 [0.00 to 10.24]
  Week 20 | 13.77 [9.47 to 18.06] | 27.20 [21.68 to 32.72] | 8.82 [0.00 to 18.36] | 13.04 [3.31 to 22.78]
  Week 28 | 19.43 [14.50 to 24.37] | 32.00 [26.22 to 37.78] | 5.88 [0.00 to 13.79] | 17.39 [6.44 to 28.34]
  Week 40 | 18.22 [13.40 to 23.03] | 30.40 [24.70 to 36.10] | 29.41 [14.10 to 44.73] | 26.09 [13.40 to 38.78]
  Week 52 | 15.79 [11.24 to 20.34] | 28.80 [23.19 to 34.41] | 29.41 [14.10 to 44.73] | 28.26 [15.25 to 41.27]

35. Secondary Outcome: Itch Severity Item (ISI) Score
Description: ISI assessed severity of itch (pruritus) due to psoriasis. ISI is a single item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends for post baseline time points. Baseline ISI is average of scores on 7 days prior to start of study treatment.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
units on a scale
  Baseline (n=343,341,62,58) | 5.49 (2.81) | 5.59 (2.72) | 5.64 (2.65) | 5.94 (2.94)
  Week 2 (n=357,358,66,64) | 3.74 (2.51) | 3.32 (2.56) | 5.45 (2.87) | 5.61 (3.04)
  Week 4 (n=351,350,64,66) | 2.89 (2.44) | 2.41 (2.28) | 5.36 (2.86) | 5.56 (3.05)
  Week 8 (n=347,348,65,66) | 2.56 (2.60) | 1.87 (2.20) | 5.51 (2.94) | 5.50 (3.35)
  Week 12 (n=343,344,65,66) | 2.38 (2.66) | 1.62 (2.18) | 4.83 (3.11) | 5.42 (3.30)
  Week 16 (n=322,335,66,66) | 2.44 (2.70) | 1.48 (2.14) | 4.82 (3.11) | 5.83 (3.27)
  Week 20 (n=312,319,66,65) | 1.94 (2.20) | 1.43 (2.23) | 2.48 (2.27) | 2.48 (2.63)
  Week 28 (n=293,306,61,61) | 1.96 (2.41) | 1.41 (2.11) | 2.02 (2.31) | 1.62 (2.09)
  Week 40 (n=202,242,53,47) | 1.47 (2.15) | 1.01 (1.77) | 1.43 (2.03) | 0.83 (1.54)
  Week 52 (n=179,218,47,46) | 1.35 (2.00) | 0.83 (1.53) | 1.60 (2.09) | 0.93 (1.44)

36. Secondary Outcome: Change From Baseline in Itch Severity Item (ISI) Score at Week 2, 4, 8, 12, 16, 20, 28, 40 and 52
Description: ISI assessed severity of itch (pruritus) due to psoriasis. ISI is a single item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo, CP-690,550 10 mg: Participants who were re-assigned to this group from placebo at Week 16 and thereafter received CP-690,550 5 mg tablet orally twice daily up to Week 52.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 340 | 339 | 62 | 58
units on a scale
  Change at Week 2 | -1.76 (0.10) | -2.25 (0.11) | -0.13 (0.25) | -0.06 (0.26)
  Change at Week 4 | -2.62 (0.11) | -3.16 (0.11) | -0.27 (0.26) | -0.11 (0.27)
  Change at Week 8 | -2.95 (0.13) | -3.72 (0.13) | -0.01 (0.29) | -0.18 (0.30)
  Change at Week 12 | -3.02 (0.13) | -3.91 (0.13) | -0.79 (0.30) | -0.25 (0.31)
  Change at Week 16 | -2.85 (0.14) | -3.97 (0.14) | -0.77 (0.31) | 0.17 (0.32)
  Change at Week 20 | -3.31 (0.13) | -3.98 (0.13) | -3.11 (0.29) | -3.16 (0.30)
  Change at Week 28 | -3.25 (0.14) | -3.94 (0.13) | -3.59 (0.30) | -4.16 (0.32)
  Change at Week 40 | -3.07 (0.15) | -3.88 (0.14) | -3.84 (0.32) | -4.40 (0.34)
  Change at Week 52 | -3.05 (0.15) | -3.89 (0.14) | -3.50 (0.32) | -4.17 (0.33)

37. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score
Description: as for outcome 5
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
units on a scale
  Baseline (n=363,359,66,66) | 12.46 (6.89) | 12.87 (6.91) | 13.83 (6.97) | 14.68 (6.80)
  Week 2 (n=356,357,66,64) | 8.65 (6.11) | 8.32 (6.45) | 11.44 (7.02) | 12.67 (7.06)
  Week 4 (n=351,349,65,66) | 6.98 (5.97) | 6.50 (5.94) | 11.45 (6.87) | 13.05 (7.14)
  Week 8 (n=345,347,65,66) | 5.88 (6.00) | 4.95 (5.58) | 10.89 (6.23) | 13.05 (7.49)
  Week 12 (n=340,344,65,66) | 5.36 (6.06) | 4.17 (5.10) | 10.29 (6.82) | 13.06 (7.58)
  Week 16 (n=319,331,66,66) | 5.45 (6.07) | 3.85 (5.17) | 10.05 (6.23) | 12.83 (7.80)
  Week 20 (n=310,319,66,65) | 4.28 (5.18) | 3.26 (4.67) | 5.89 (4.88) | 7.17 (6.69)
  Week 28 (n=289,303,61,61) | 3.94 (5.05) | 3.24 (4.83) | 4.34 (4.88) | 3.46 (4.27)
  Week 40 (n=200,239,53,46) | 2.53 (4.11) | 2.11 (3.79) | 3.25 (4.43) | 1.63 (2.17)
  Week 52 (n=177,216,47,46) | 2.86 (4.35) | 1.91 (3.72) | 3.40 (4.43) | 1.78 (2.44)

38. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 2, 4, 8, 12, 16, 20, 28, 40 and 52
Description: as for outcome 5
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 358 | 357 | 66 | 66
units on a scale
  Change at Week 2 | -4.02 (0.23) | -4.56 (0.23) | -1.94 (0.54) | -1.07 (0.54)
  Change at Week 4 | -5.65 (0.25) | -6.41 (0.25) | -1.90 (0.57) | -0.77 (0.57)
  Change at Week 8 | -6.68 (0.27) | -7.95 (0.27) | -2.45 (0.61) | -0.77 (0.61)
  Change at Week 12 | -7.09 (0.27) | -8.70 (0.27) | -3.08 (0.63) | -0.75 (0.63)
  Change at Week 16 | -6.97 (0.29) | -8.90 (0.28) | -3.33 (0.65) | -0.98 (0.65)
  Change at Week 20 | -8.01 (0.27) | -9.42 (0.27) | -7.48 (0.61) | -6.48 (0.61)
  Change at Week 28 | -8.25 (0.28) | -9.36 (0.28) | -9.02 (0.62) | -9.72 (0.62)
  Change at Week 40 | -8.50 (0.30) | -9.51 (0.29) | -9.26 (0.63) | -10.89 (0.65)
  Change at Week 52 | -8.26 (0.31) | -9.56 (0.30) | -9.23 (0.65) | -10.90 (0.66)

39. Secondary Outcome: 36-Item Short-Form Health Survey Version 2, Acute (SF-36)
Description: 36-Item Short-Form Health Survey (SF-36) is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects are summarized as physical and mental health summary scores. The score range for the physical and mental health scores is 0-100 (100=highest level of functioning).
Time Frame: Baseline, Week 16, 28, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
units on a scale
  Baseline: Physical Health Score (n=358,355,66,66) | 47.36 (9.10) | 47.02 (9.05) | 47.12 (8.95) | 44.86 (9.12)
  Baseline: Mental Health Score (n=358,355,66,66) | 42.98 (12.53) | 43.35 (11.57) | 42.53 (11.77) | 42.97 (11.44)
  Week 16: Physical Health Score (n=318,329,65,65) | 49.83 (8.34) | 50.99 (8.63) | 48.04 (8.75) | 45.60 (8.87)
  Week 16: Mental Health Score (n=318,329,65,65) | 47.23 (10.93) | 49.06 (9.50) | 44.47 (10.77) | 43.07 (12.34)
  Week 28: Physical Health Score (n=286,303,60,61) | 51.01 (7.67) | 51.92 (7.86) | 51.11 (8.08) | 49.63 (8.52)
  Week 28: Mental Health Score (n=286,303,60,61) | 48.59 (10.47) | 49.64 (9.35) | 48.63 (9.57) | 49.69 (9.71)
  Week 52: Physical Health Score (n=177,216,46,46) | 51.98 (7.10) | 52.42 (7.93) | 50.90 (8.75) | 52.12 (7.64)
  Week 52: Mental Health Score (n=177,216,46,46) | 49.05 (10.33) | 50.73 (8.38) | 50.77 (9.43) | 49.58 (9.67)

40. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Score
Description: HADS: 14-item questionnaire that screens for the presence of anxiety and depression symptoms. There are 7 items comprising the anxiety subscale, and 7 items comprising the depression subscale. Each item has response option ranging from 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score ranges from 0 to 21 for each subscale; higher score indicates greater severity of anxiety or depression symptoms.
Time Frame: Baseline, Week 4, 16, 28, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
units on a scale
  Baseline: Anxiety Subscale (n=362,358,66,66) | 6.58 (4.21) | 6.21 (4.08) | 6.94 (4.21) | 7.06 (4.02)
  Baseline: Depression Subscale (n=362,358,66,66) | 5.20 (4.27) | 5.09 (4.09) | 5.61 (3.98) | 5.68 (3.93)
  Week 4: Anxiety Subscale (n=350,349,65,66) | 5.66 (3.96) | 5.30 (3.90) | 6.82 (4.11) | 6.70 (4.12)
  Week 4: Depression Subscale (n=350,349,65,66) | 4.34 (3.59) | 4.23 (3.75) | 5.28 (4.06) | 5.26 (4.12)
  Week 16: Anxiety Subscale (n=317,333,65,66) | 5.50 (4.18) | 4.74 (3.76) | 6.20 (4.39) | 6.85 (4.50)
  Week 16: Depression Subscale (n=317,333,65,66) | 3.97 (3.87) | 3.51 (3.71) | 4.92 (3.65) | 5.50 (4.07)
  Week 28: Anxiety Subscale (n=286,304,60,61) | 4.98 (4.04) | 4.47 (4.00) | 4.60 (3.89) | 4.82 (3.88)
  Week 28: Depression Subscale (n=286,304,60,61) | 3.63 (3.64) | 3.21 (3.65) | 3.65 (3.66) | 3.59 (3.25)
  Week 52: Anxiety Subscale (n=177,215,46,46) | 3.97 (3.65) | 3.84 (3.88) | 4.33 (4.21) | 4.00 (3.81)
  Week 52:Depression Subscale (n= 177, 215, 46, 46) | 3.05 (3.48) | 2.80 (3.49) | 3.11 (3.16) | 3.09 (3.03)

41. Secondary Outcome: Work Limitation Questionnaire (WLQ) Index Score
Description: WLQ: participant-reported 25-item scale to evaluate degree to which health problems interfere with an ability to perform job roles along 4 dimensions: Time Management scale (5 items); Physical Demands scale (6 items); Mental-Interpersonal Demands Scale (9 items); Output Demands Scale (5 items). All the scales ranged from 0 (limited none of the time) to 100 (limited all of the time). The WLQ Index score is the weighted sum of the scores from the 4 WLQ scales (total score: 0 [no loss] to 100 [complete loss of work]).
Time Frame: Baseline, Week 4, 16, 28, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
units on a scale
  Baseline (n= 309, 305, 55, 56) | 7.40 (6.38) | 7.90 (6.51) | 7.16 (5.84) | 8.40 (6.01)
  Week 4 (n= 291, 298, 53, 55) | 6.92 (6.68) | 6.64 (6.42) | 6.67 (6.41) | 9.66 (6.55)
  Week 16 (n= 273, 279, 51, 55) | 6.68 (6.37) | 5.72 (5.93) | 6.53 (5.97) | 7.13 (5.69)
  Week 28 (n= 241, 254, 51, 53) | 6.12 (6.37) | 5.77 (6.29) | 6.03 (6.29) | 6.24 (6.36)
  Week 52 (n= 148, 183, 41, 41) | 6.02 (6.26) | 5.95 (6.65) | 6.73 (6.54) | 5.29 (6.49)

42. Secondary Outcome: Percentage of Participants With Patient Global Assessment (PtGA) Scale Response
Description: The PtGA asks the participant to evaluate the overall cutaneous disease at that point in time on a single item, 5-point scale (0=clear [no psoriasis]; 1=almost clear; 2=mild; 3=moderate; 4=severe).
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
percentage of participants
  Baseline: Clear (n = 360, 359, 66, 66) | 0.0 | 0.0 | 0.0 | 0.0
  Baseline: Almost Clear (n = 360, 359, 66, 66) | 0.0 | 0.0 | 0.0 | 0.0
  Baseline: Mild (n = 360, 359, 66, 66) | 1.9 | 3.6 | 3.0 | 1.5
  Baseline: Moderate (n = 360, 359, 66, 66) | 35.3 | 35.7 | 31.8 | 34.8
  Baseline: Severe (n = 360, 359, 66, 66) | 62.8 | 60.7 | 65.2 | 63.6
  Week 2: Clear (n = 357, 358, 66, 64) | 0.0 | 0.3 | 0.0 | 0.0
  Week 2: Almost Clear (n = 357, 358, 66, 64) | 1.1 | 3.9 | 0.0 | 0.0
  Week 2: Mild (n = 357, 358, 66, 64) | 14.8 | 17.6 | 7.6 | 6.3
  Week 2: Moderate (n = 357, 358, 66, 64) | 51.0 | 48.0 | 37.9 | 40.6
  Week 2: Severe (n = 357, 358, 66, 64) | 33.1 | 30.2 | 54.5 | 53.1
  Week 4: Clear (n = 350, 348, 65, 65) | 0.0 | 0.9 | 0.0 | 0.0
  Week 4: Almost Clear (n = 350, 348, 65, 65) | 10.0 | 12.1 | 1.5 | 0.0
  Week 4: Mild (n = 350, 348, 65, 65) | 24.6 | 29.9 | 7.7 | 4.6
  Week 4: Moderate (n = 350, 348, 65, 65) | 42.9 | 40.5 | 46.2 | 36.9
  Week 4: Severe (n = 350, 348, 65, 65) | 22.6 | 16.7 | 44.6 | 58.5
  Week 8: Clear (n = 345, 346, 65, 66) | 1.7 | 3.8 | 0.0 | 0.0
  Week 8: Almost Clear (n = 345, 346, 65, 66) | 19.7 | 27.7 | 1.5 | 1.5
  Week 8: Mild (n = 345, 346, 65, 66) | 29.3 | 28.9 | 12.3 | 6.1
  Week 8: Moderate (n = 345, 346, 65, 66) | 30.1 | 27.2 | 43.1 | 39.4
  Week 8: Severe (n = 345, 346, 65, 66) | 19.1 | 12.4 | 43.1 | 53.0
  Week 12: Clear (n = 341, 344, 65, 65) | 3.8 | 8.7 | 0.0 | 0.0
  Week 12: Almost Clear (n = 341, 344, 65, 65) | 24.9 | 35.2 | 3.1 | 3.1
  Week 12: Mild (n = 341, 344, 65, 65) | 29.6 | 27.9 | 23.1 | 7.7
  Week 12: Moderate (n = 341, 344, 65, 65) | 24.3 | 19.5 | 32.3 | 33.8
  Week 12: Severe (n = 341, 344, 65, 65) | 17.3 | 8.7 | 41.5 | 55.4
  Week 16: Clear (n = 320, 331, 66, 66) | 3.4 | 10.9 | 0.0 | 0.0
  Week 16: Almost Clear (n = 320, 331, 66, 66) | 28.4 | 37.8 | 6.1 | 3.0
  Week 16: Mild (n = 320, 331, 66, 66) | 30.6 | 24.8 | 15.2 | 10.6
  Week 16: Moderate (n = 320, 331, 66, 66) | 22.5 | 19.0 | 42.4 | 25.8
  Week 16: Severe (n = 320, 331, 66, 66) | 15.0 | 7.6 | 36.4 | 60.6
  Week 20: Clear (n = 311, 319, 65, 64) | 6.1 | 16.3 | 0.0 | 1.6
  Week 20: Almost Clear (n = 311, 319, 65, 64) | 34.1 | 35.7 | 23.1 | 20.3
  Week 20: Mild (n = 311, 319, 65, 64) | 28.6 | 27.3 | 26.2 | 20.3
  Week 20: Moderate (n = 311, 319, 65, 64) | 23.5 | 13.5 | 46.2 | 35.9
  Week 20: Severe (n = 311, 319, 65, 64) | 7.7 | 7.2 | 4.6 | 21.9
  Week 28: Clear (n = 290, 303, 61, 61) | 11.7 | 20.8 | 6.6 | 14.8
  Week 28: Almost Clear (n = 290, 303, 61, 61) | 36.9 | 40.6 | 32.8 | 39.3
  Week 28: Mild (n = 290, 303, 61, 61) | 19.3 | 17.5 | 39.3 | 29.5
  Week 28: Moderate (n = 290, 303, 61, 61) | 25.2 | 15.8 | 19.7 | 11.5
  Week 28: Severe (n = 290, 303, 61, 61) | 6.9 | 5.3 | 1.6 | 4.9
  Week 40: Clear (n = 200, 239, 53, 46) | 18.5 | 30.5 | 11.3 | 28.3
  Week 40: Almost Clear (n = 200, 239, 53, 46) | 44.0 | 41.4 | 50.9 | 56.5
  Week 40: Mild (n = 200, 239, 53, 46) | 18.5 | 15.5 | 20.8 | 15.2
  Week 40: Moderate (n = 200, 239, 53, 46) | 16.0 | 11.3 | 15.1 | 0.0
  Week 40: Severe (n = 200, 239, 53, 46) | 3.0 | 1.3 | 1.9 | 0.0
  Week 52: Clear (n = 177, 216, 47, 46) | 14.1 | 32.9 | 19.1 | 34.8
  Week 52: Almost Clear (n = 177, 216, 47, 46) | 45.8 | 39.8 | 31.9 | 45.7
  Week 52: Mild (n = 177, 216, 47, 46) | 17.5 | 15.3 | 23.4 | 13.0
  Week 52: Moderate (n = 177, 216, 47, 46) | 16.4 | 9.3 | 21.3 | 6.5
  Week 52: Severe (n = 177, 216, 47, 46) | 6.2 | 2.8 | 4.3 | 0.0

43. Secondary Outcome: Percentage of Participants With Patient Satisfaction With Study Medication (PSSM) Score Response
Description: The PSSM is a single, 7 point item that evaluates overall participant satisfaction with the study treatment. Response options range from "very dissatisfied" to "very satisfied" with the study treatment.
Time Frame: Week 16, 28, 52
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
percentage of participants
  Week16:Not Satisfied/Dissatisfied(n=317,332,65,66) | 6.0 | 6.3 | 12.3 | 13.6
  Week 16:Slightly Dissatisfied (n=317,332,65,66) | 3.2 | 1.5 | 9.2 | 7.6
  Week 16:Slightly Satisfied (n=317,332,65,66) | 7.9 | 6.9 | 9.2 | 12.1
  Week 16:Somewhat Dissatisfied (n=317,332,65,66) | 6.0 | 3.0 | 9.2 | 18.2
  Week 16:Somewhat Satisfied (n=317,332,65,66) | 22.1 | 22.9 | 16.9 | 7.6
  Week 16:Very Dissatisfied (n=317,332,65,66) | 5.4 | 4.2 | 29.2 | 33.3
  Week 16:Very Satisfied (n=317,332,65,66) | 49.5 | 55.1 | 13.8 | 7.6
  Week28:Not Satisfied/Dissatisfied(n=285,303,60,61) | 2.1 | 4.0 | 1.7 | 3.3
  Week 28:Slightly Dissatisfied (n=285,303,60,61) | 4.6 | 3.3 | 1.7 | 1.6
  Week 28:Slightly Satisfied (n=285,303,60,61) | 10.5 | 6.9 | 11.7 | 3.3
  Week 28:Somewhat Dissatisfied (n=285,303,60,61) | 3.9 | 0.7 | 0.0 | 1.6
  Week 28:Somewhat Satisfied (n=285,303,60,61) | 27.0 | 26.1 | 40.0 | 31.1
  Week 28:Very Dissatisfied (n=285,303,60,61) | 2.5 | 3.6 | 0.0 | 0.0
  Week 28:Very Satisfied (n=285,303,60,61) | 49.5 | 55.4 | 45.0 | 59.0
  Week52:Not Satisfied/Dissatisfied(n=176,217,46,46) | 2.8 | 0.9 | 0.0 | 0.0
  Week 52:Slightly Dissatisfied (n=176,217,46,46) | 1.1 | 0.9 | 2.2 | 0.0
  Week 52:Slightly Satisfied (n=176,217,46,46) | 5.1 | 5.5 | 13.0 | 0.0
  Week 52:Somewhat Dissatisfied (n=176,217,46,46) | 2.3 | 0.9 | 2.2 | 0.0
  Week 52:Somewhat Satisfied (n=176,217,46,46) | 33.5 | 25.3 | 34.8 | 28.3
  Week 52:Very Dissatisfied (n=176,217,46,46) | 0.0 | 0.9 | 0.0 | 0.0
  Week 52:Very Satisfied (n=176,217,46,46) | 55.1 | 65.4 | 47.8 | 71.7

44. Secondary Outcome: Joint Pain Assessment (JPA) Score
Description: The JPA assesses severity of joint pain. The JPA is a horizontal numeric rating scale. Participants were asked to "select the number that best describes any joint pain that participant may have experienced over the past 24 hours" with response options ranging from "0-no joint pain" to "10-worst possible joint pain."
Time Frame: Baseline, Week 4, 16, 28, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
units on a scale
  Baseline (n= 363, 359, 66, 65) | 3.42 (3.21) | 2.96 (2.99) | 3.00 (2.94) | 3.69 (3.15)
  Week 4 (n= 351, 349, 64, 66) | 2.24 (2.57) | 2.13 (2.56) | 3.13 (2.68) | 3.18 (3.19)
  Week 16 (n= 319, 333, 65, 66) | 2.41 (2.76) | 1.89 (2.59) | 3.20 (3.07) | 3.45 (3.22)
  Week 28 (n= 287, 304, 60, 60) | 2.08 (2.53) | 1.71 (2.46) | 1.93 (2.18) | 1.93 (2.36)
  Week 52 (n= 176, 215, 46, 46) | 1.60 (2.25) | 1.38 (2.25) | 1.46 (2.24) | 1.50 (2.41)

45. Secondary Outcome: Euro Quality of Life 5 Dimensions (EQ-5D) - Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Week 16, 28, 40, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
units on a scale
  Baseline (n= 363, 359, 66, 65) | 0.77 (0.19) | 0.77 (0.19) | 0.78 (0.17) | 0.74 (0.19)
  Week 16 (n= 319, 333, 65, 65) | 0.86 (0.16) | 0.88 (0.15) | 0.81 (0.18) | 0.76 (0.19)
  Week 28 (n= 288, 303, 60, 61) | 0.86 (0.15) | 0.89 (0.14) | 0.89 (0.14) | 0.88 (0.13)
  Week 40 (n= 201, 239, 53, 46) | 0.91 (0.13) | 0.91 (0.15) | 0.92 (0.14) | 0.90 (0.16)
  Week 52 (n= 176, 217, 47, 46) | 0.89 (0.12) | 0.90 (0.14) | 0.89 (0.14) | 0.90 (0.13)

46. Secondary Outcome: Euro Quality of Life 5 Dimensions (EQ-5D) - Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 millimeter (mm) (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Week 16, 28, 40, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 363 | 360 | 66 | 66
mm
  Baseline (n= 361, 359, 65, 66) | 67.28 (22.53) | 66.97 (22.63) | 68.65 (21.20) | 65.24 (19.61)
  Week 16 (n= 316, 330, 64, 66) | 76.00 (18.96) | 77.95 (17.36) | 69.00 (17.95) | 59.85 (22.92)
  Week 28 (n= 287, 303, 60, 61) | 77.99 (17.89) | 78.89 (17.38) | 76.37 (18.10) | 79.13 (12.80)
  Week 40 (n= 201, 240, 53, 46) | 81.47 (17.74) | 83.84 (15.09) | 82.96 (12.25) | 83.80 (12.62)
  Week 52 (n= 175, 216, 47, 45) | 80.23 (17.42) | 84.59 (13.80) | 81.23 (14.54) | 82.38 (13.73)

47. Secondary Outcome: Psoriasis Healthcare Resource Utilization Questionnaire (Ps-HCRU) - Interaction With Healthcare Professional
Description: The Psoriasis Health Care Resource Utilization (Ps-HCRU) questionnaire is a short questionnaire designed to assess healthcare resource use and the impact of psoriasis on work. The first section assesses direct costs associated with healthcare resource use (interactions with healthcare providers such as general practitioners, Dermatologist, Rheumatologist). Baseline is the latest pre-dose measurement. Week 16 includes all reported log data to Week 16 (excluding Baseline). Participants may have response in more than 1 category. Data was not analyzed beyond Week 16 as per study team's decision because Week 0 - 16 period was considered sufficient to provide clear reflection of Ps-HCRU endpoint.
Time Frame: Baseline, Week 16
Population: FAS included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (CP-690,550 or placebo). Here 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies participants evaluable at specified time point for each arm, respectively.
Measure: Number; unit: events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 56 | 57 | 23
events
  Baseline: General Practitioner (n= 28, 39, 15) | 3 | 5 | 2
  Baseline: Dermatologist (n= 28, 39, 15) | 24 | 34 | 14
  Baseline: Rheumatologist (n= 28, 39, 15) | 0 | 1 | 0
  Baseline: Cardiologist (n= 28, 39, 15) | 0 | 1 | 0
  Baseline: Gastroenterologist (n= 28, 39, 15) | 0 | 0 | 0
  Baseline: Psychiatrist (n= 28, 39, 15) | 0 | 0 | 0
  Baseline: Surgeon (n= 28, 39, 15) | 0 | 0 | 0
  Baseline: Nurse (n= 28, 39, 15) | 9 | 5 | 3
  Baseline: Other (n= 28, 39, 15) | 1 | 2 | 1
  Week 16: General Practitioner (n= 56, 57, 23) | 33 | 32 | 12
  Week 16: Dermatologist (n= 56, 57, 23) | 14 | 22 | 8
  Week 16: Rheumatologist (n= 56, 57, 23) | 0 | 0 | 0
  Week 16: Cardiologist (n= 56, 57, 23) | 1 | 0 | 1
  Week 16: Gastroenterologist (n= 56, 57, 23) | 0 | 0 | 2
  Week 16: Psychiatrist (n= 56, 57, 23) | 2 | 3 | 0
  Week 16: Surgeon (n= 56, 57, 23) | 4 | 3 | 1
  Week 16: Nurse (n= 56, 57, 23) | 2 | 4 | 2
  Week 16: Other (n= 56, 57, 23) | 23 | 18 | 7

48. Secondary Outcome: Psoriasis Healthcare Resource Utilization Questionnaire (Ps-HCRU) - Impact of Psoriasis on Work
Description: The Psoriasis Health Care Resource Utilization (Ps-HCRU) questionnaire is a short questionnaire designed to assess healthcare resource use and the impact of psoriasis on work. The second section assesses indirect costs associated with absenteeism due to psoriasis and the impact of psoriasis on productivity at work. Participants employed at the time of assessment answered (Yes/No [Y/N]): "Were you absent or on sick leave from work due to psoriasis today?", and participants unemployed (UEmp) at the time of assessment answered (Yes/No): "Are you unemployed due to your psoriasis?" Baseline is the latest pre-dose measurement. Week 16 includes all reported log up to Week 16 (excluding Baseline). Data was not analyzed beyond Week 16 as per study team's decision because Week 0 - 16 period was considered sufficient to provide clear reflection of Ps-HCRU endpoint.
Time Frame: Baseline, Week 16
Population: FAS included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (CP-690,550 or placebo). Here 'n' signifies those participants who were evaluable for this measure at specified time point for each arm, respectively.
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 363 | 360 | 177
participants
  Baseline: Emp, Absent/Sick Leave:Y (n=237,232,114) | 55 | 47 | 27
  Baseline: Emp, Absent/Sick Leave:N (n=237,232,114) | 182 | 185 | 87
  Baseline: UEmp, due to Psoriasis:Y (n=97,103,49) | 15 | 24 | 4
  Baseline: UEmp, due to Psoriasis:N (n=97,103,49) | 82 | 79 | 45
  Week 16: Emp, Absent/Sick Leave:Y (n=224,221,88) | 47 | 37 | 24
  Week 16: Emp, Absent/Sick Leave:N (n=224,221,88) | 177 | 184 | 64
  Week 16: UEmp, due to Psoriasis:Y (n=77,87,42) | 10 | 13 | 6
  Week 16:UEmp, due to Psoriasis: N (n=77,87,42) | 67 | 74 | 36

49. Secondary Outcome: Psoriasis Healthcare Resource Utilization Questionnaire (Ps-HCRU) - Healthcare Resource Use Events and Employment Status
Description: The Psoriasis Health Care Resource Utilization (Ps-HCRU) questionnaire is a short questionnaire designed to assess healthcare resource use and the impact of psoriasis on work. The first section assesses direct costs associated with healthcare resource use, and the second section assesses indirect costs associated with absenteeism due to psoriasis and the impact of psoriasis on productivity at work. Percentage of participants reporting healthcare resource use events and employment status, work impacted events due to psoriasis, and absence or sick leave for work due to psoriasis at Week 16 are reported. Data was not analyzed beyond Week 16 as per study team's decision because Week 0 - 16 period was considered sufficient to provide clear reflection of Ps-HCRU endpoint.
Time Frame: Week 16
Population: FAS included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (CP-690,550 or placebo). Here 'n' signifies those participants who were evaluable (answered respective question for this measure) for specified parameter for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 363 | 360 | 177
percentage of participants
  Healthcare Resource Use Events (n=30,37,5) | 100.00 | 94.59 | 100.00
  Employment (n=301,310,130) | 74.42 | 71.94 | 66.92
  Work Impacted Events (n=79,88,42) | 12.66 | 14.77 | 14.29
  Absence/Sick Leave Due to Psoriasis (n=224,221,90) | 20.98 | 16.74 | 27.78

50. Secondary Outcome: Psoriasis Healthcare Resource Utilization Questionnaire (Ps-HCRU) - Work Hours and Absent Hours
Description: The Psoriasis Health Care Resource Utilization (Ps-HCRU) questionnaire is a short questionnaire designed to assess healthcare resource use and the impact of psoriasis on work. The first section assesses direct costs associated with healthcare resource use, and the second section assesses indirect costs associated with absenteeism due to psoriasis and the impact of psoriasis on productivity at work. Baseline is the latest pre-dose measurement. Participants reported hours scheduled to work and hours absent from work. Data was not analyzed beyond Week 16 as per study team's decision because Week 0 - 16 period was considered sufficient to provide clear reflection of Ps-HCRU endpoint.
Time Frame: Baseline, Week 16
Population: FAS included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (CP-690,550 or placebo). Here 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies participants evaluable for specified parameter for each arm, respectively.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 54 | 48 | 27
hours
  Baseline: Hours Scheduled to Work (n=54,48,25) | 8.61 (1.31) | 8.15 (1.75) | 7.92 (0.91)
  Baseline: Hours Absent From Work (n=54,47,27) | 5.15 (3.09) | 6.00 (3.03) | 5.81 (2.48)
  Week 16: Hours Scheduled to Work (n=47,39,25) | 8.49 (1.80) | 8.31 (1.08) | 8.40 (1.63)
  Week 16: Hours Absent From Work (n=46,38,24) | 5.41 (3.15) | 5.24 (2.39) | 5.88 (2.40)

51. Secondary Outcome: Psoriasis Healthcare Resource Utilization Questionnaire (Ps-HCRU) - Percent Absent Hours
Description: The Psoriasis Health Care Resource Utilization (Ps-HCRU) questionnaire is a short questionnaire designed to assess healthcare resource use and the impact of psoriasis on work. The first section assesses direct costs associated with healthcare resource use, and the second section assesses indirect costs associated with absenteeism due to psoriasis and the impact of psoriasis on productivity at work. Baseline is the latest pre-dose measurement. Participants reported hours scheduled to work and hours absent from work. Percent absent hours = (hours absent from work/hours scheduled to work) multiplied by 100. Data was not analyzed beyond Week 16 as per study team's decision because Week 0 - 16 period was considered sufficient to provide clear reflection of Ps-HCRU endpoint.
Time Frame: Baseline, Week 16
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: percentage of scheduled hours
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 53 | 47 | 25
percentage of scheduled hours
  Baseline (n=53,47,25) | 60.32 (33.29) | 72.84 (32.96) | 75.76 (30.04)
  Week 16 (n=46,38,24) | 64.15 (35.08) | 65.21 (31.55) | 71.81 (30.99)

52. Secondary Outcome: Psoriasis Healthcare Resource Utilization Questionnaire (Ps-HCRU) - Psoriasis Affecting Ability to Work
Description: The Psoriasis Health Care Resource Utilization (Ps-HCRU) questionnaire is a short questionnaire designed to assess healthcare resource use and the impact of psoriasis on work. The first section assesses direct costs associated with healthcare resource use, and the second section assesses indirect costs associated with absenteeism due to psoriasis and the impact of psoriasis on productivity at work. Baseline is the latest pre-dose measurement. Participants rate how much psoriasis affected their ability to work by reporting a number from 0 to 10, where 0 means "ability to work was not affected by psoriasis", and 10 means "ability to work was completely affected by psoriasis". Data was not analyzed beyond Week 16 as per study team's decision because Week 0 - 16 period was considered sufficient to provide clear reflection of Ps-HCRU endpoint.
Time Frame: Baseline, Week 16
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 363 | 360 | 177
units on a scale
  Baseline (n=238,234,114) | 2.23 (2.81) | 2.13 (2.64) | 2.89 (3.07)
  Week 16 (n=223,222,89) | 1.13 (2.13) | 1.26 (2.60) | 1.94 (2.53)

53. Secondary Outcome: Family Dermatology Life Quality Index (FDLQI) Score
Description: The FDLQI is a 10-item questionnaire that examine the impact of health-related quality of life issues associated with living with a person with a skin condition (example, emotional distress, personal relationships, reactions of other people, social life, caregiving) over the last month. The FDLQI need to be completed by a family member (for example, spouse or partner, parent) who currently lives with the participant. Each question is scored on a scale from 0 (Not at all/ Not relevant) to 3 (Very much). Total score is calculated by summing the score of each item resulting in a maximum score of '30' and a minimum score of '0'. Higher scores indicate greater impairment to quality of life.
Time Frame: Baseline, Week 16, 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg
Number analyzed (Participants) | 22 | 27 | 5 | 5
units on a scale
  Baseline (n= 22, 27, 5, 5) | 9.45 (7.40) | 9.41 (7.45) | 9.40 (3.78) | 8.80 (3.03)
  Week 16 (n= 17, 17, 5, 5) | 3.76 (4.25) | 3.53 (4.16) | 6.20 (5.26) | 6.40 (4.28)
  Week 52 (n= 6, 9, 3, 2) | 1.17 (2.40) | 2.00 (4.21) | 5.67 (3.51) | 0.50 (0.71)

ADVERSE EVENTS:
Description: Same event may appear as both AE/SAE; distinct events are presented. An event may be categorized as serious in 1 subject and as nonserious in another subject, or 1 subject may have experienced both a serious and nonserious event during the study. Adverse events for participants (n=45) who were not re-randomized at week 16, are reported separately.
Groups:
- Placebo, CP-690,550 5 mg: Placebo matched to CP-690,550 tablet orally twice daily up to Week 16 and thereafter CP-690,550 5 mg tablet orally twice daily up to Week 52.
- Placebo, CP-690,550 10 mg: Placebo matched to CP-690,550 tablet orally twice daily up to Week 16 and thereafter CP-690,550 10 mg tablet orally twice daily up to Week 52.
- Placebo: Participants who received placebo matched to CP-690,550 tablet orally twice daily up to Week 16 but were not re-randomized to CP-690,550 treatment.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, CP-690,550 5 mg | Placebo, CP-690,550 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 24/363 | 19/360 | 1/66 | 6/66 | 2/45
Other Adverse Events (participants affected / at risk) | 189/363 | 222/360 | 44/66 | 38/66 | 22/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg (N=363) | CP-690,550 10 mg (N=360) | Placebo, CP-690,550 5 mg (N=66) | Placebo, CP-690,550 10 mg (N=66) | Placebo (N=45)
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pelvic mass (General disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Burn infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Mycobacterium test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg (N=363) | CP-690,550 10 mg (N=360) | Placebo, CP-690,550 5 mg (N=66) | Placebo, CP-690,550 10 mg (N=66) | Placebo (N=45)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 4 | 2 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 0 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 8 | 2 | 1 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 13 | 2 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 5 | 1 | 0 | 2
Food poisoning (Gastrointestinal disorders) | 3 | 1 | 2 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 12 | 13 | 1 | 5 | 0
Toothache (Gastrointestinal disorders) | 4 | 9 | 0 | 0 | 0
Chest pain (General disorders) | 3 | 3 | 0 | 0 | 1
Fatigue (General disorders) | 8 | 6 | 1 | 1 | 2
Hyperthermia (General disorders) | 2 | 3 | 2 | 1 | 0
Oedema peripheral (General disorders) | 3 | 2 | 0 | 1 | 1
Pain (General disorders) | 0 | 2 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1 | 1 | 1 | 1
Folliculitis (Infections and infestations) | 2 | 8 | 1 | 3 | 0
Gastroenteritis (Infections and infestations) | 2 | 9 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 6 | 3 | 1 | 0
Herpes zoster (Infections and infestations) | 4 | 8 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 11 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 38 | 55 | 11 | 9 | 4
Oral herpes (Infections and infestations) | 4 | 4 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 4 | 4 | 3 | 2 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 3 | 2 | 1 | 0
Rhinitis (Infections and infestations) | 4 | 4 | 2 | 2 | 0
Sinusitis (Infections and infestations) | 7 | 5 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 33 | 35 | 4 | 4 | 0
Urinary tract infection (Infections and infestations) | 12 | 12 | 5 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 3 | 2 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 4 | 2 | 1 | 0 | 1
Bacterial test positive (Investigations) | 0 | 1 | 3 | 0 | 0
Blood cholesterol increased (Investigations) | 9 | 13 | 2 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 26 | 38 | 3 | 7 | 0
Blood triglycerides increased (Investigations) | 6 | 5 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 8 | 9 | 0 | 4 | 0
Haemoglobin decreased (Investigations) | 2 | 2 | 2 | 0 | 0
Low density lipoprotein increased (Investigations) | 10 | 10 | 1 | 2 | 0
Gout (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 15 | 17 | 1 | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 10 | 18 | 1 | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 2 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 11 | 5 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 6 | 2 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 4 | 0 | 2 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 3 | 1 | 0
Dizziness (Nervous system disorders) | 7 | 4 | 2 | 0 | 0
Headache (Nervous system disorders) | 28 | 28 | 4 | 3 | 0
Insomnia (Psychiatric disorders) | 2 | 3 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 2 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 5 | 9 | 1 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 9 | 4 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.